CLINICAL TRIAL: NCT01587703
Title: A Phase I/II Open-Label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GSK525762 in Subjects With NUT Midline Carcinoma (NMC) and Other Cancers
Brief Title: A Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GSK525762 in Subjects With NUT Midline Carcinoma (NMC) and Other Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115521; 2014-004982-25 (EudraCT Number)
Record Dates: First submitted 2012-04-03; First posted 2012-04-30 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Midline
Keywords: BRD3; GSK525762; NUT Midline Carcinoma; MYCN-amplified Solid Tumor; BRD4; BET inhibitor; bromodomains; NMC; Colorectal C ancer; Small Cell Lung Cancer; Multiple Myeloma; Neuroblastoma; Oncology
MeSH Terms: conditions — Carcinoma; Small Cell Lung Carcinoma; Multiple Myeloma; Neuroblastoma; Neoplasms | interventions — molibresib

ARMS (3):
- Single and Repeat Dose finding cohort (Experimental): All subjects will follow a 3+3 dose escalation design for GSK525762 and the dose will be escalated based on all available data, including PK data and the safety profile of prior cohorts, as well as the recommended dose from the Neuenschwander- Continuous Reassessment Method (N-CRM) design.
  Interventions: Drug: GSK525762
- Expansion Cohort (Experimental): Up to 150 additional subjects with NMC and other solid tumors may be enrolled in expansion cohorts. The recommended Phase 2 (Part 2) dose (RP2D) of GSK525762 will be determined based on the MTD or biologically active dose (example: clinical response), the safety profile and available pharmacodynamic data generated from all subjects in Parts 1
  Interventions: Drug: GSK525762
- Besylate Sub study (Experimental): Tablet and amorphous tablet in one of the two sequences (ABCD or BACD). Where Treatment A: RP2D/MTD as amorphous free-base tablet + low dose stable isotope in solution, fasted Treatment B: RP2D/MTD as besylate tablet + low dose stable isotope in solution, fasted. Treatment C: half to one-third of RP2D/MTD as besylate tablet + low dose stable isotope in solution, fasted. Treatment D: RP2D/MTD as besylate tablet, fed
  Interventions: Drug: GSK525762

INTERVENTIONS:
Drug: GSK525762 — Begin at Dose Level 1 and increase up to 2 fold

SUMMARY:
This study is divided into two parts; Part 1 of the study is a dose escalation phase to select the recommended dose for Part 2 based on the safety, pharmacokinetic, and pharmacodynamic profiles observed after oral administration of GSK525762 in the following subjects: NMC, small cell lung cancer (SCLC), non-small cell lung cancer (NSCLC), colorectal cancer (CRC), neuroblastoma (NB), castration resistant prostate cancer (CRPC), triple negative breast cancer (TNBC), estrogen receptor positive (ER positive) breast cancer, and MYCN driven solid tumor subjects. Part 2 of the study will explore the safety, tolerability, pharmacokinetics, pharmacodynamics, and clinical activity of the recommended dose from Part 1 in cohorts comprised of NMC, small cell lung cancer (SCLC), castration resistant prostate cancer (CRPC), triple negative breast cancer (TNBC), and estrogen receptor positive (ER positive) breast cancer subjects. Approximately 60 subjects will be enrolled in the Part 1 and approximately 150 subjects will be enrolled in Part 2. A sub-study will be opened in Part 1 to approximately 10-12 subjects in the United States to investigate the relative bioavailability of the besylate tablet compared to the amorphous free-base tablet at the maximum tolerated dose (MTD) or recommended phase 2 dosing (RP2D), the effect of high-fat high-calorie meal on the bioavailability of the besylate tablet at the MTD or RP2D and the dose proportionality of 2 doses of GSK525762 administered as besylate tablet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 16 years or older, at the time of signing the informed consent.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. If the subject is less than 18 years old, an Assent form and parental/guardian Consent form (replacing "you will" with "your child will" will be required).
* Diagnosis of one of the following: Part 1 Only: NUT Midline Carcinoma based on ectopic expression of NUT protein as determined by IHC and/or detection of NUT gene translocation as determined by FISH. Subjects may be treatment naïve or have had prior therapy; SCLC, CRC, NB, TNBC, ER positive BC, CRPC, NSCLC and any other solid tumor which has been confirmed by clinical testing to be MYCN amplified (defined as a MYCN gene copy number gain of >=5). Subjects should have tumor progression after receiving at least one prior standard/approved chemotherapy, or where there is no approved therapy, or where standard therapy is refused. Part 2 only: NUT Midline Carcinoma as diagnosed by the Central Laboratory. Subjects may be treatment naïve or have had prior therapy. SCLC, CRPC, TNBC and ER+BC .
* Subjects with solid tumors, with the exception of CRPC, must demonstrate measurable disease, per RECIST v1.1. NOTE: Subjects with NMC that do not meet the RECIST v1.1 criteria for measurable disease, but have evaluable disease may be considered for enrollment after discussion with the GSK medical monitor..
* All prior treatment- related toxicities must be CTCAE (Version 4.0) <=Grade 1 (except alopecia and peripheral neuropathy) at the time of treatment allocation [NCI-CTCAE, 2009].
* ECOG Performance Status score of 0 or 2 for subjects with NMC; 0-1 for subjects with other tumor types.
* Adequate organ function as follows: Hematologic system: Absolute neutrophil count (ANC), Lab values - >=1.5 X 10^9/L; Hematologic system: Hemoglobin, Lab values - >=9.5 grams/deciliter (g/dL) (subjects that required transfusion or growth factor need to demonstrate stable haemoglobin for 7 days of 9.5 g/ g/dL); Hematologic system: Platelets, Lab values - >=100 X 10^9/Liter [L] ); Hematologic system: Prothrombin time /International normalized ratio and partial thromboplastin time, Lab values - <=1.5 X upper limit of normal (ULN). Renal system: Creatinine, lab values - <=1.5 X ULN; or Renal system: Calculated creatinine clearance [calculated by Cockcroft Gault formula], lab values - >=50 milliliter (mL)/minute (min); or Renal system: 24-hour urine creatinine clearance>=50 mL/min; Hepatic system: total Bilirubin <=1.5 X ULN (isolated bilirubin >1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin <35% or subject has a diagnosis of Gilbert's syndrome), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >=2.5 x ULN. Cardiac system: Ejection fraction, lab values - >=lower limit of normal (LLN) by Echocardiogram (ECHO) (minimum of 50%); Cardiac system: Troponin ( T), lab values - <=ULN; Cardiac system: Potassium, lab values - >=LLN and <=ULN; Cardiac system: Magnesium, lab values - >=LLN. Thyroid system: thyroid stimulating hormone, lab values >=LLN and <=to ULN. Reproductive /endocrine system: testosterone <50 nanogram (ng)/dL (only for subject with CRPC)
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 milli international unit/mL and estradiol less than 40 pg/mL (less than 140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential and agrees to use one of the contraception methods (described in the protocol) for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 7 months after the last dose of study medication; Negative serum pregnancy test <=7 days prior to first study drug dose; Female subjects who are lactating must discontinue nursing prior to the first dose of study treatment and must refrain from nursing throughout the treatment period and for 5 half-lives of GSK525762 or at least 28 days (whichever is longer) following the last dose of study treatment.
* Male subjects must agree to use one of the methods of contraception specified. This method must be used from the time of the first dose of study medication until least 16 weeks after the last dose of study medication. In addition, male subjects whose partners are or become pregnant while on study medication must continue to use condoms for 7 days after stopping study medications.
* Specific eligibility criteria for Part 2 CRPC expansion cohort: Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma, surgically castrated or continuously medically castrated (for >=8 weeks prior to pre-screening).
* Specific eligibility criteria for Part 2 CRPC expansion cohort: Persistent disease with evidence of disease progression following standard therapy(ies) including prior treatment with androgen/androgen receptor directed therapy, including enzalutamide and/or abiraterone
* Specific eligibility criteria for Part 2 CRPC expansion cohort: Ongoing androgen deprivation therapy with a serum testosterone level <1.7 nanomoles/L or <50 ng/dL.
* Specific eligibility criteria for Part 2 CRPC expansion cohort: Prostate-Specific Antigen (PSA) levels >=2.0 ng/mL. Note: If PSA level has been obtained within 14 days of Screening, this test does not need to be repeated and the result previously obtained may be used for the Screening value.

Exclusion Criteria:

* Primary malignancy of the central nervous system or malignancies related to human immunodeficiency virus or solid organ transplant. History of known HIV. History of known Hepatitis B surface antigen or positive Hepatitis C antibody (confirmed by RIBA).
* Prior treatments usage as defined: A) Use of an investigational anti-cancer drug within 14 days or 5 half-lives, whichever is longer, prior to the first dose of the investigational products:; B) A minimum of 14 days between termination of the investigational drug and administration of GSK525762; C) Any therapy related toxicities must also have resolved to Grade 1 or less. Note that an investigational drug is defined as a drug without an approved oncologic indication; D) Chemotherapy, radiotherapy, anti-neoplastic antibody or targeted therapy or immunotherapy within 14 days, major surgery within 28 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of the investigational product. Anti-androgen (e.g., bicalutamide) therapies for prostate cancer must be stopped 4 weeks prior to enrollment. Second line hormone therapies such as enzalutamide, abiraterone, or orteronel should be stopped 2 weeks prior to enrollment. Subjects with prostate cancer should remain on luteinizing hormone releasing hormone (LHRH) agonists or antagonists. Subjects with prostate cancer may also remain on low-dose prednisone or prednisolone (up to 10 mg/day) and still be eligible for this study.
* Current use of anticoagulants (e.g., warfarin, heparin) at therapeutic levels within 7 days prior to the first dose of GSK525762. Low dose (prophylactic) low molecular weight heparin (LMWH) is permitted. In addition, INR must be monitored in accordance with local institutional practices.
* Current use of a prohibited medication or requires any of these medications during treatment with the investigational drugs (details will be available in the protocol). This includes excluding current medications known or suspected to be associated QT prolongation. In addition, any subject who may require a QT prolonging medication while on trial should not be enrolled.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes). Any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. NOTE: Subjects previously treated for these conditions that have had stable central nervous system disease (verified with consecutive imaging studies) for >1 month, are asymptomatic and off corticosteroids, or are on stable dose of corticosteroids for at least 1 month prior to study Day 1 are permitted. Stability of brain metastases must be confirmed with imaging. Subject treated with gamma knife the can be enrolled 2 weeks post-procedure as long as there are no post-procedure complications/stable. In addition, subjects treated or currently taking enzyme-inducing anticonvulsant are allowed on study.
* Cardiac abnormalities as evidenced by any of the following: History or current "untreated" clinically significant uncontrolled arrhythmias; Clinically significant conduction abnormalities or arrhythmias, subjects with Bundle Branch Block; Presence of cardiac pacemaker; History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA); History of acute coronary syndromes (including unstable angina and myocardial infarction ), coronary angioplasty, or stenting within the past 3 months.
* Any of the following ECG findings: Baseline QTcF interval >=450 millisecond (msec); Any clinically significant ECG assessments should be reviewed by the site cardiologist prior to study entry.
* GSK525762 is a benzodiazepine class molecule. Any serious known immediate or delayed hypersensitivity reaction(s) to GSK525762 or idiosyncrasy to drugs chemically related to the investigational drug.
* Hemoptysis >1 teaspoon in 24 hours within the last 28 days.
* History of major gastrointestinal bleeding within the last 6 months. Any evidence of active gastrointestinal bleeding excludes the subject.
* Besylate Sub-Study only: unable or unwilling to eat the FDA recommended high-fat high-calorie breakfast (two eggs fried in butter, two strips of bacon, 4 ounce [oz]) of hash brown potatoes and 8 oz of whole milk) within the recommended 30 minutes.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (5):
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Clayton, Victoria, Australia
- France (3):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
- GSK Investigational Site, Amsterdam, Netherlands
- GSK Investigational Site, Seoul, South Korea
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
- United Kingdom (2):
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Background] Piha-Paul SA, Hann CL, French CA, Cousin S, Brana I, Cassier PA, Moreno V, de Bono JS, Harward SD, Ferron-Brady G, Barbash O, Wyce A, Wu Y, Horner T, Annan M, Parr NJ, Prinjha RK, Carpenter CL, Hilton J, Hong DS, Haas NB, Markowski MC, Dhar A, O'Dwyer PJ, Shapiro GI. Phase 1 Study of Molibresib (GSK525762), a Bromodomain and Extra-Terminal Domain Protein Inhibitor, in NUT Carcinoma and Other Solid Tumors. JNCI Cancer Spectr. 2019 Nov 6;4(2):pkz093. doi: 10.1093/jncics/pkz093. eCollection 2020 Apr. PMID 32328561
- [Derived] Cousin S, Blay JY, Garcia IB, de Bono JS, Le Tourneau C, Moreno V, Trigo J, Hann CL, Azad AA, Im SA, Cassier PA, French CA, Italiano A, Keedy VL, Plummer R, Sablin MP, Hemming ML, Ferron-Brady G, Wyce A, Khaled A, Datta A, Foley SW, McCabe MT, Wu Y, Horner T, Kremer BE, Dhar A, O'Dwyer PJ, Shapiro GI, Piha-Paul SA. Safety, pharmacokinetic, pharmacodynamic and clinical activity of molibresib for the treatment of nuclear protein in testis carcinoma and other cancers: Results of a Phase I/II open-label, dose escalation study. Int J Cancer. 2022 Mar 15;150(6):993-1006. doi: 10.1002/ijc.33861. Epub 2021 Nov 26. PMID 34724226
- [Derived] Krishnatry AS, Voelkner A, Dhar A, Prohn M, Ferron-Brady G. Population pharmacokinetic modeling of molibresib and its active metabolites in patients with solid tumors: A semimechanistic autoinduction model. CPT Pharmacometrics Syst Pharmacol. 2021 Jul;10(7):709-722. doi: 10.1002/psp4.12639. Epub 2021 Jun 4. PMID 33955700
- [Derived] Parikh SA, French CA, Costello BA, Marks RS, Dronca RS, Nerby CL, Roden AC, Peddareddigari VG, Hilton J, Shapiro GI, Molina JR. NUT midline carcinoma: an aggressive intrathoracic neoplasm. J Thorac Oncol. 2013 Oct;8(10):1335-8. doi: 10.1097/JTO.0b013e3182a00f41. PMID 24457244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 196 participants were enrolled and randomized in the Part 1 QD (65 participants), Part 1 BID (19 participants), Besylate Substudy (10 participants), and Part 2 (102 participants) groups.
Pre-assignment Details: This was a 2-Part study conducted in 8 countries-Part 1 (dose-escalation) and Part 2 (dose expansion). A besylate sub-study (four period, crossover) was conducted in 10 participants in the United States.
Groups:
- Part 1: GSK525762 2 mg QD: Participants were administered once daily (QD) oral dose of 2 milligrams (mg) GSK525762.
- Part 1: GSK525762 4 mg QD: Participants were administered once daily oral dose of 4 mg GSK525762
- Part 1: GSK525762 8 mg QD: Participants were administered once daily oral dose of 8 mg GSK525762.
- Part 1: GSK525762 16 mg QD: Participants were administered once daily oral dose of 16 mg GSK525762.
- Part 1: GSK525762 30 mg QD: Participants were administered once daily oral dose of 30 mg GSK525762.
- Part 1: GSK525762 60 mg QD: Participants were administered once daily oral dose of 60 mg GSK525762.
- Part 1: GSK525762 80 mg QD: Participants were administered once daily oral dose of 80 mg GSK525762.
- Part 1: GSK525762 100 mg QD: Participants were administered once daily oral dose of 100 mg GSK525762.
- Part 1: GSK525762 20 mg BID: Participants were administered twice daily (BID) oral dose of 20 mg GSK525762.
- Part 1: GSK525762 30 mg BID: Participants were administered twice daily oral dose of 30 mg GSK525762.
- Part 1: GSK525762 40 mg BID: Participants were administered twice daily oral dose of 40 mg GSK525762.
- Part 2: Participants With NMC: Participants with NUT Midline Carcinoma (NMC) were administered continuous once daily oral dose of 75 mg GSK525762.
- Part 2: Participants With SCLC: Participants with small cell lung cancer(SCLC) were administered continuous once daily oral dose of 75 mg GSK525762
- Part 2: Participants With CRPC: Participants with Castrate-Resistant Prostate Cancer (CRPR) were administered continuous once daily oral dose of 75 mg GSK525762
- Part 2: Participants With TNBC: Participants with Triple Negative Breast Cancer (TNBC) were administered continuous once daily oral dose of 75 mg GSK525762.
- Part 2: Participants With ER+BC: Participants with estrogen receptor positive breast cancer (ER+BC) were administered continuous once daily oral dose of 75 mg GSK525762
- Part 2: Participants With GIST: Participants with Gastrointestinal Stromal Tumor (GIST) were administered continuous once daily oral dose of 75 mg GSK525762.
- 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes: Participants received GSK525762 80 mg amorphous (amor) free-base tablet along with 6 mg stable isotope (iso) in solution in the fasted state in Period 1 followed by administration of GSK525762 80 mg besylate (bes) tablet along with 6 mg stable iso in solution in the fasted state in Period 2. Participants were then administered GSK525762 30 mg bes tablet along with 6 mg stable iso in solution in the fasted state in Period 3 and GSK525762 80 mg bes tablet was administered with Food and Drug Administration (FDA) recommended high fat breakfast in Period 4.
- 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes: Participants received GSK525762 80 mg bes tablet along with 6 mg stable iso in solution in the fasted state in Period 1 followed by administration GSK525762 80 mg amor free-base tablet along with 6 mg stable iso in solution in the fasted state in Period 2. Participants were then administered GSK525762 30 mg bes tablet along with 6 mg stable iso in solution in the fasted state in Period 3 and GSK525762 80 mg bes tablet was administered with FDA recommended high fat breakfast in Period 4.
Period: Part1 QD(Median Exposure of 1.38months)
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Started | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 1 | 3 | 4 | 8 | 32 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site closed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 4 | 1 | 3 | 4 | 7 | 30 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part1 BID(Median Exposure of 1.41months)
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 10 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy-Period(P)1, Week1(Day1 to Day3)
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy-P2, Week1Day3 to Week2Day1
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy-P3, Week2Day1 to Week2Day3
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy-P4,Maximum Exposure of 5.5month
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4
Period: Part2(Median Exposure of 1.41 Months)
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 14 | 23 | 19 | 21 | 13 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 14 | 22 | 19 | 21 | 13 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Site closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 3 | 8 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 12 | 21 | 16 | 17 | 5 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants in Besylate Substudy: All participants who entered besylate sub-study and received 80 mg amor free-base tablet along with 6 mg stable iso in solution in fasted state; 80 mg bes tablet along with 6 mg stable iso in solution in fasted state, 30 mg bes tablet along with 6 mg stable iso in solution in fasted state and 80 mg bes tablet with FDA recommended high fat breakfast in one of the treatment periods were included.
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | All Participants in Besylate Substudy | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 1: GSK525762 2 mg QD | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | Total
Number analyzed (Participants) | 4 | 1 | 3 | 4 | 9 | 32 | 9 | 4 | 10 | 5 | 10 | 12 | 14 | 23 | 3 | 19 | 21 | 13 | 196
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (19.44) | 39.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed | 53.7 (4.19) | 49.3 (23.27) | 46.7 (17.06) | 51.5 (16.82) | 58.3 (19.92) | 66.5 (6.45) | 63.5 (8.42) | 60.4 (4.83) | 55.2 (9.96) | 42.9 (18.05) | 58.3 (11.04) | 63.8 (6.11) | 40.0 (15.77) | 50.8 (8.66) | 59.7 (10.34) | 61.0 (13.23) | 55.4 (14.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 6 | 14 | 2 | 2 | 4 | 1 | 5 | 7 | 9 | 0 | 1 | 19 | 21 | 6 | 105
  Male | 1 | 0 | 0 | 3 | 3 | 18 | 7 | 2 | 6 | 4 | 5 | 5 | 5 | 23 | 2 | 0 | 0 | 7 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Central/South Asian Heritage (Her) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Japanese Her/East Asian Her/South East Asian Her | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 9
  Black or African American | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 12
  White | 3 | 0 | 2 | 4 | 7 | 30 | 8 | 3 | 10 | 5 | 9 | 6 | 8 | 23 | 2 | 15 | 18 | 10 | 163
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 2 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Part 1 QD
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the outcomes mentioned; events of possible study treatment-induced liver injury with hyperbilirubinemia; any new primary cancers; significant cardiac dysfunction; Grade 4 laboratory abnormalities; and drug related hepatobiliary event leading to permanent discontinuation of study treatment. All Treated Population comprised of all participants who received at least one dose of study treatment.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants
  Any AE | 3 | 4 | 1 | 3 | 3 | 9 | 31 | 9
  Any SAE | 0 | 2 | 0 | 0 | 1 | 2 | 21 | 3

2. Primary Outcome: Number of Participants With AEs and SAEs-Part 1 BID
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the outcomes mentioned; events of possible study treatment-induced liver injury with hyperbilirubinemia; any new primary cancers; significant cardiac dysfunction; Grade 4 laboratory abnormalities; and drug related hepatobiliary event leading to permanent discontinuation of study treatment
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  Any AE | 4 | 10 | 5
  Any SAE | 0 | 4 | 2

3. Primary Outcome: Number of Participants With AEs and SAEs-Part 2
Description: as for outcome 2
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Groups:
- Participants With NMC: Participants with NUT Midline Carcinoma (NMC) were administered continuous once daily oral dose of 75 mg GSK525762
- Participants With SCLC: Participants with small cell lung cancer(SCLC) were administered continuous once daily oral dose of 75 mg GSK525762
- Participants With CRPC: Participants with Castrate-Resistant Prostate Cancer (CRPC) were administered continuous once daily oral dose of 75 mg GSK525762
- Participants With TNBC: Participants with Triple Negative Breast Cancer (TNBC) were administered continuous once daily oral dose of 75 mg GSK525762
- Participants With ER+BC: Participants with estrogen receptor positive breast cancer (ER+BC) were administered continuous once daily oral dose of 75 mg GSK525762
- Participants With GIST: Participants with Gastrointestinal Stromal Tumor (GIST) were administered continuous once daily oral dose of 75 mg GSK525762
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Participants
  Any AE | 11 | 14 | 23 | 19 | 21 | 13
  Any SAE | 6 | 9 | 16 | 11 | 15 | 8

4. Primary Outcome: Number of Participants With Dose Reductions or Delays-Part 1 QD
Description: The number of participants who had any dose reductions or delays is presented.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 7

5. Primary Outcome: Number of Participants With Dose Reductions or Delays-Part 1 BID
Description: The number of participants who had any dose reductions or delays is presented.
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants | 0 | 3 | 1

6. Primary Outcome: Number of Participants With Dose Reductions or Delays-Part 2
Description: The number of participants who had any dose reductions or delays is presented.
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Participants | 7 | 4 | 11 | 6 | 6 | 4

7. Primary Outcome: Number of Participants With Dose Reductions or Delays-Besylate Sub-study
Description: The number of participants who had any dose reductions or delays is presented.
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants | 3 | 1

8. Primary Outcome: Number of Participants Withdrawn Due to Toxicities-Part 1 QD
Description: Number of participants withdrawn due to toxicities is presented.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants | 0 | 1 | 0 | 0 | 0 | 2 | 7 | 2

9. Primary Outcome: Number of Participants Withdrawn Due to Toxicities-Part 1 BID
Description: Number of participants withdrawn due to toxicities is presented.
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants | 0 | 2 | 2

10. Primary Outcome: Number of Participants Withdrawn Due to Toxicities-Part 2
Description: Number of participants withdrawn due to toxicities is presented.
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Participants | 1 | 3 | 6 | 4 | 6 | 2

11. Primary Outcome: Number of Participants Withdrawn Due to Toxicities-Besylate Sub-study
Description: Number of participants withdrawn due to toxicities is presented.
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

12. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Part 1 QD
Description: Blood samples were collected for the analysis of: glucose, albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), amylase, aspartate aminotransferase (AST), direct bilirubin (Dir bil), bilirubin, N-Terminal proB-type natriuretic peptide (NT-BNP), calcium, cholesterol, creatine kinase (CK), chloride, carbon dioxide (CO2), creatinine, gamma glutamyl transferase (GGT), high and low density lipoprotein (HDL and LDL), insulin, potassium, lactate dehydrogenase (LDH), lipase, magnesium, protein, sodium, thyroxine, testosterone, triglycerides, troponin I and T, urate and urea. Grading was done according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death. Baseline is the most recent, non-missing value prior to or on first study treatment dose date. Data for worst case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.38 months of drug exposure
Population: All Treated Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants
  Glucose; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Glucose; Any grade increase; n=2,4,1,3,4,9,32,9 | 0 | 2 | 1 | 3 | 2 | 7 | 24 | 8
  Glucose; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Glucose; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Glucose; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Glucose; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Albumin; Any grade increase; n=2,4,1,3,4,9,32,9 | 0 | 2 | 0 | 0 | 1 | 3 | 12 | 1
  Albumin; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Albumin; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Albumin; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP; Any grade increase; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  ALP; Any grade increase; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0
  ALP; Increase to Grade 3; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  ALP; Increase to Grade 3; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALP; Increase to Grade 4; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  ALP; Increase to Grade 4; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  ALT; Any grade increase; n=2,4,1,3,4,9,32,9 | 0 | 0 | 1 | 0 | 1 | 1 | 9 | 2
  ALT; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  ALT; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  ALT; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Amylase; Any grade increase; n=2,4,1,3,4,9,32,9 | 1 | 1 | 0 | 1 | 2 | 0 | 10 | 1
  Amylase; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Amylase; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Amylase; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Amylase; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  AST; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  AST; Any grade increase; n=2,4,1,3,4,9,32,9 | 2 | 1 | 1 | 0 | 2 | 1 | 14 | 3
  AST; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  AST; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AST; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  AST; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dir bil; Any grade increase; n=2,4,1,3,4,9,30,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 30 | 9
  Dir bil; Any grade increase; n=2,4,1,3,4,9,30,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dir bil; Increase to Grade 3; n=2,4,1,3,4,9,30,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 30 | 9
  Dir bil; Increase to Grade 3; n=2,4,1,3,4,9,30,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dir bil; Increase to Grade 4; n=2,4,1,3,4,9,30,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 30 | 9
  Dir bil; Increase to Grade 4; n=2,4,1,3,4,9,30,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Bilirubin; Any grade increase; n=2,4,1,3,4,9,32,9 | 0 | 0 | 1 | 0 | 1 | 1 | 15 | 8
  Bilirubin; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Bilirubin; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 1
  Bilirubin; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Bilirubin; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NT-BNP; Any grade increase; n=2,4,1,3,4,9,30,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 30 | 9
  NT-BNP; Any grade increase; n=2,4,1,3,4,9,30,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NT-BNP; Increase to Grade 3; n=2,4,1,3,4,9,30,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 30 | 9
  NT-BNP; Increase to Grade 3; n=2,4,1,3,4,9,30,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NT-BNP; Increase to Grade 4; n=2,4,1,3,4,9,30,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 30 | 9
  NT-BNP; Increase to Grade 4; n=2,4,1,3,4,9,30,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Calcium; Any grade increase; n=2,4,1,3,4,9,32,9 | 1 | 1 | 0 | 1 | 2 | 1 | 17 | 3
  Calcium; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Calcium; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Calcium; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cholesterol;Any grade increase;n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Cholesterol;Any grade increase;n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 1
  Cholesterol;Increase to Grade 3;n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Cholesterol;Increase to Grade 3;n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cholesterol;Increase to Grade 4;n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Cholesterol;Increase to Grade 4;n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CK;Any grade increase;n=3,4,1,3,4,9,31,9: number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  CK;Any grade increase;n=3,4,1,3,4,9,31,9 | 0 | 1 | 0 | 0 | 1 | 0 | 11 | 5
  CK; Increase to Grade 3; n=3, 4, 1, 3, 4, 9, 31, 9: number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  CK; Increase to Grade 3; n=3, 4, 1, 3, 4, 9, 31, 9 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  CK; Increase to Grade 4; n=3, 4, 1, 3, 4, 9, 31, 9: number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  CK; Increase to Grade 4; n=3, 4, 1, 3, 4, 9, 31, 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride; Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Chloride; Any grade increase; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride; Increase to Grade 3;n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Chloride; Increase to Grade 3;n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride;Increase to Grade 4;n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Chloride;Increase to Grade 4;n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CO2; Any grade increase; n=2, 4, 1, 3, 4, 9, 32, 9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  CO2; Any grade increase; n=2, 4, 1, 3, 4, 9, 32, 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CO2; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  CO2; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CO2; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  CO2; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine;Any grade increase;n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Creatinine;Any grade increase;n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 3
  Creatinine;Increase to Grade 3;n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Creatinine;Increase to Grade 3;n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine;Increase to Grade 4;n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Creatinine;Increase to Grade 4;n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT; Any grade increase; n=2, 4, 1, 3, 4, 9, 31, 7: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 7
  GGT; Any grade increase; n=2, 4, 1, 3, 4, 9, 31, 7 | 0 | 1 | 0 | 0 | 1 | 0 | 11 | 1
  GGT;Increase to Grade 3; n=2,4,1,3,4,9,31,7: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 7
  GGT;Increase to Grade 3; n=2,4,1,3,4,9,31,7 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  GGT; Increase to Grade 4; n=2,4,1,3,4,9,31,7: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 7
  GGT; Increase to Grade 4; n=2,4,1,3,4,9,31,7 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HDL; Any grade increase; n=2, 4, 1, 3, 4, 7, 28, 9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 28 | 9
  HDL; Any grade increase; n=2, 4, 1, 3, 4, 7, 28, 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HDL; Increase to Grade 3; n=2,4,1,3,4,7,28,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 28 | 9
  HDL; Increase to Grade 3; n=2,4,1,3,4,7,28,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HDL; Increase to Grade 4; n=2,4,1,3,4,7,28,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 28 | 9
  HDL; Increase to Grade 4; n=2,4,1,3,4,7,28,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Insulin; Any grade increase; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Insulin; Any grade increase; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Insulin; Increase to Grade 3; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Insulin; Increase to Grade 3; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Insulin; Increase to Grade 4; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Insulin; Increase to Grade 4; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium;Any grade increase;n=3,4,1,3,4,9,32,9 | 2 | 2 | 0 | 3 | 0 | 2 | 13 | 3
  Potassium;Increase to Grade 3;n=3,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Potassium;Increase to Grade 4;n=3,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  LDH; Any grade increase; n=0, 0, 0, 0, 0, 1, 0, 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LDH; Any grade increase; n=0, 0, 0, 0, 0, 1, 0, 0 |  |  |  |  |  | 0 |  |
  LDH; Increase to Grade 3; n=0, 0, 0, 0, 0, 1, 0, 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LDH; Increase to Grade 3; n=0, 0, 0, 0, 0, 1, 0, 0 |  |  |  |  |  | 0 |  |
  LDH; Increase to Grade 4; n=0, 0, 0, 0, 0, 1, 0, 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LDH; Increase to Grade 4; n=0, 0, 0, 0, 0, 1, 0, 0 |  |  |  |  |  | 0 |  |
  LDL; Any grade increase; n=2, 4, 1, 3, 4, 7, 28, 8: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 28 | 8
  LDL; Any grade increase; n=2, 4, 1, 3, 4, 7, 28, 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LDL;Increase to Grade 3; n=2,4,1,3,4,7,28,8: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 28 | 8
  LDL;Increase to Grade 3; n=2,4,1,3,4,7,28,8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LDL;Increase to Grade 4; n=2,4,1,3,4,7,28,8: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 28 | 8
  LDL;Increase to Grade 4; n=2,4,1,3,4,7,28,8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase;Any grade increase; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Lipase;Any grade increase; n=2,4,1,3,4,9,31,9 | 1 | 0 | 0 | 0 | 0 | 0 | 8 | 2
  Lipase;Increase to Grade 3; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Lipase;Increase to Grade 3; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Lipase;Increase to Grade 4; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Lipase;Increase to Grade 4; n=2,4,1,3,4,9,31,9 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Magnesium;Any grade increase;n=3,4,1,3,4,9,32,9 | 0 | 2 | 1 | 1 | 1 | 0 | 9 | 2
  Magnesium;Increase to Grade 3;n=3,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Magnesium;Increase to Grade 4;n=3,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein;Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Protein;Any grade increase; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein;Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Protein;Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein;Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Protein;Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium;Any grade increase; n=3,4,1,3,4,9,32,9 | 1 | 3 | 0 | 1 | 2 | 3 | 16 | 4
  Sodium;Increase to Grade 3; n=3,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
  Sodium;Increase to Grade 4; n=3,4,1,3,4,9,32,9 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Thyroxine;Any grade increase;n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Thyroxine;Any grade increase;n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Thyroxine;Increase to Grade 3; n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Thyroxine;Increase to Grade 3; n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Thyroxine;Increase to Grade 4; n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Thyroxine;Increase to Grade 4; n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Testosterone;Any grade increase;n=1,0,0,0,3,3,14,7: number analyzed (Participants) | 1 | 0 | 0 | 0 | 3 | 3 | 14 | 7
  Testosterone;Any grade increase;n=1,0,0,0,3,3,14,7 | 0 |  |  |  | 0 | 0 | 0 | 0
  Testosterone;Increase to Grade3;n=1,0,0,0,3,3,14,7: number analyzed (Participants) | 1 | 0 | 0 | 0 | 3 | 3 | 14 | 7
  Testosterone;Increase to Grade3;n=1,0,0,0,3,3,14,7 | 0 |  |  |  | 0 | 0 | 0 | 0
  Testosterone;Increase to Grade4;n=1,0,0,0,3,3,14,7: number analyzed (Participants) | 1 | 0 | 0 | 0 | 3 | 3 | 14 | 7
  Testosterone;Increase to Grade4;n=1,0,0,0,3,3,14,7 | 0 |  |  |  | 0 | 0 | 0 | 0
  Triglyc;Any grade increase;n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Triglyc;Any grade increase;n=2,4,1,3,4,7,29,9 | 0 | 2 | 0 | 0 | 2 | 2 | 17 | 6
  Triglyc;Increase to Grade 3;n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Triglyc;Increase to Grade 3;n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Triglyc;Increase to Grade 4;n=2,4,1,3,4,7,29,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 7 | 29 | 9
  Triglyc;Increase to Grade 4;n=2,4,1,3,4,7,29,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Troponin I;Any grade increase;n=0,0,0,0, 2,5,24,5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 5 | 24 | 5
  Troponin I;Any grade increase;n=0,0,0,0, 2,5,24,5 |  |  |  |  | 0 | 0 | 0 | 0
  Troponin I;Increase to Grade 3;n=0,0,0,0,2,5,24,5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 5 | 24 | 5
  Troponin I;Increase to Grade 3;n=0,0,0,0,2,5,24,5 |  |  |  |  | 0 | 0 | 0 | 0
  Troponin I;Increase to Grade 4; n=0,0,0,0,2,5,24,5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 5 | 24 | 5
  Troponin I;Increase to Grade 4; n=0,0,0,0,2,5,24,5 |  |  |  |  | 0 | 0 | 0 | 0
  Troponin T;Any grade increase;n=3,4,1,3,4,9,31,9: number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Troponin T;Any grade increase;n=3,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin T;Increase to Grade 3; n=3,4,1,3,4,9,31,9: number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Troponin T;Increase to Grade 3; n=3,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin T;Increase to Grade 4; n=3,4,1,3,4,9,31,9: number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Troponin T;Increase to Grade 4; n=3,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urate;Any grade increase; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Urate;Any grade increase; n=2,4,1,3,4,9,32,9 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Urate; Increase to Grade 3; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Urate; Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urate; Increase to Grade 4; n=2,4,1,3,4,9,32,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
  Urate; Increase to Grade 4; n=2,4,1,3,4,9,32,9 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Urea; Any grade increase; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Urea; Any grade increase; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea; Increase to Grade 3; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Urea; Increase to Grade 3; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea; Increase to Grade 4; n=2,4,1,3,4,9,31,9: number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 31 | 9
  Urea; Increase to Grade 4; n=2,4,1,3,4,9,31,9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Part 1 BID
Description: Blood samples were collected for the analysis of clinical chemistry parameters: glucose, albumin, ALP, ALT, amylase, AST, Dir bil, bilirubin, NT-BNP, calcium, cholesterol, CK, chloride, CO2, creatinine, GGT, HDL and LDL cholesterol, insulin, potassium, LDH, lipase, magnesium, protein, sodium, thyroxine, testosterone, triglycerides, troponin I and T, urate and urea. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: GSK525762 20 mg BID: Participants were administered twice daily oral dose of 20 mg GSK525762.
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  Glucose; Any grade increase; n=4, 10, 5 | 1 | 9 | 5
  Glucose; Increase to Grade 3; n=4, 10, 5 | 1 | 3 | 1
  Glucose; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Albumin; Any grade increase; n=4, 10, 5 | 0 | 4 | 1
  Albumin; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Albumin; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  ALP; Any grade increase; n=4, 10, 5 | 0 | 4 | 2
  ALP; Increase to Grade 3; n=4, 10, 5 | 0 | 2 | 0
  ALP; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  ALT; Any grade increase; n=4, 10, 5 | 0 | 5 | 1
  ALT; Increase to Grade 3; n=4, 10, 5 | 0 | 1 | 0
  ALT; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Amylase; Any grade increase; n=4, 10, 5 | 0 | 2 | 2
  Amylase; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Amylase; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  AST; Any grade increase; n=4, 10, 5 | 2 | 6 | 1
  AST; Increase to Grade 3; n=4, 10, 5 | 0 | 2 | 0
  AST; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Dir bil; Any grade increase; n=4, 9, 4: number analyzed (Participants) | 4 | 9 | 4
  Dir bil; Any grade increase; n=4, 9, 4 | 0 | 0 | 0
  Dir bil; Increase to Grade 3; n=4, 9, 4: number analyzed (Participants) | 4 | 9 | 4
  Dir bil; Increase to Grade 3; n=4, 9, 4 | 0 | 0 | 0
  Dir bil; Increase to Grade 4; n=4, 9, 4: number analyzed (Participants) | 4 | 9 | 4
  Dir bil; Increase to Grade 4; n=4, 9, 4 | 0 | 0 | 0
  Bilirubin; Any grade increase; n=4, 10, 5 | 1 | 7 | 2
  Bilirubin; Increase to Grade 3; n=4, 10, 5 | 1 | 1 | 1
  Bilirubin; Increase to Grade 4; n=4, 10, 5 | 0 | 1 | 0
  NT-BNP; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  NT-BNP; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  NT-BNP; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Calcium; Any grade increase; n=4, 10, 5 | 1 | 2 | 1
  Calcium; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Calcium; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Cholesterol; Any grade increase; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  Cholesterol; Any grade increase; n=2, 9, 5 | 0 | 2 | 0
  Cholesterol; Increase to Grade 3; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  Cholesterol; Increase to Grade 3; n=2, 9, 5 | 0 | 0 | 0
  Cholesterol; Increase to Grade 4; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  Cholesterol; Increase to Grade 4; n=2, 9, 5 | 0 | 0 | 0
  CK; Any grade increase; n=4, 10, 5 | 0 | 3 | 2
  CK; Increase to Grade 3; n=n=4, 10, 5 | 0 | 0 | 0
  CK; Increase to Grade 4; n=n=4, 10, 5 | 0 | 0 | 0
  Chloride; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  Chloride; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Chloride; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  CO2; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  CO2; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  CO2; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Creatinine; Any grade increase; n=4, 10, 5 | 0 | 2 | 2
  Creatinine; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Creatinine; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  GGT; Any grade increase; n=4, 10, 5 | 0 | 4 | 1
  GGT; Increase to Grade 3; n=4, 10, 5 | 0 | 1 | 0
  GGT; Increase to Grade 4; n=4, 10, 5 | 0 | 1 | 0
  HDL; Any grade increase; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  HDL; Any grade increase; n=2, 9, 5 | 0 | 0 | 0
  HDL; Increase to Grade 3; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  HDL; Increase to Grade 3; n=2, 9, 5 | 0 | 0 | 0
  HDL; Increase to Grade 4; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  HDL; Increase to Grade 4; n=2, 9, 5 | 0 | 0 | 0
  Insulin; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  Insulin; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Insulin; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Potassium; Any grade increase; n=4, 10, 5 | 1 | 5 | 2
  Potassium; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Potassium; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  LDL; Any grade increase; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  LDL; Any grade increase; n=2, 9, 5 | 0 | 0 | 0
  LDL; Increase to Grade 3; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  LDL; Increase to Grade 3; n=2, 9, 5 | 0 | 0 | 0
  LDL; Increase to Grade 4; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  LDL; Increase to Grade 4; n=2, 9, 5 | 0 | 0 | 0
  Lipase; Any grade increase; n=4, 10, 5 | 0 | 2 | 3
  Lipase; Increase to Grade 3; n=4, 10, 5 | 0 | 1 | 0
  Lipase; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Magnesium; Any grade increase; n=4, 10, 5 | 0 | 2 | 2
  Magnesium; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Magnesium; Increase to Grade 4; n=4, 10, 5 | 0 | 1 | 0
  Protein; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  Protein; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Protein; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Sodium; Any grade increase; n=4, 10, 5 | 0 | 7 | 2
  Sodium; Increase to Grade 3; n=4, 10, 5 | 0 | 2 | 0
  Sodium; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Thyroxine; Any grade increase; n=3, 9, 5: number analyzed (Participants) | 3 | 9 | 5
  Thyroxine; Any grade increase; n=3, 9, 5 | 0 | 0 | 0
  Thyroxine; Increase to Grade 3; n=3, 9, 5: number analyzed (Participants) | 3 | 9 | 5
  Thyroxine; Increase to Grade 3; n=3, 9, 5 | 0 | 0 | 0
  Thyroxine; Increase to Grade 4; n=3, 9, 5: number analyzed (Participants) | 3 | 9 | 5
  Thyroxine; Increase to Grade 4; n=3, 9, 5 | 0 | 0 | 0
  Testosterone; Any grade increase; n=1, 4, 4: number analyzed (Participants) | 1 | 4 | 4
  Testosterone; Any grade increase; n=1, 4, 4 | 0 | 0 | 0
  Testosterone; Increase to Grade 3; n=1, 4, 4: number analyzed (Participants) | 1 | 4 | 4
  Testosterone; Increase to Grade 3; n=1, 4, 4 | 0 | 0 | 0
  Testosterone; Increase to Grade 4; n=1, 4, 4: number analyzed (Participants) | 1 | 4 | 4
  Testosterone; Increase to Grade 4; n=1, 4, 4 | 0 | 0 | 0
  Triglycerides; Any grade increase; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  Triglycerides; Any grade increase; n=2, 9, 5 | 0 | 4 | 4
  Triglycerides; Increase to Grade 3; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  Triglycerides; Increase to Grade 3; n=2, 9, 5 | 0 | 0 | 0
  Triglycerides; Increase to Grade 4; n=2, 9, 5: number analyzed (Participants) | 2 | 9 | 5
  Triglycerides; Increase to Grade 4; n=2, 9, 5 | 0 | 0 | 0
  Troponin I; Any grade increase; n=3, 10, 5: number analyzed (Participants) | 3 | 10 | 5
  Troponin I; Any grade increase; n=3, 10, 5 | 0 | 0 | 0
  Troponin I; Increase to Grade 3; n=3, 10, 5: number analyzed (Participants) | 3 | 10 | 5
  Troponin I; Increase to Grade 3; n=3, 10, 5 | 0 | 0 | 0
  Troponin I; Increase to Grade 4; n=3, 10, 5: number analyzed (Participants) | 3 | 10 | 5
  Troponin I; Increase to Grade 4; n=3, 10, 5 | 0 | 0 | 0
  Troponin T; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  Troponin T; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Troponin T; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Urate; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  Urate; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Urate; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0
  Urea; Any grade increase; n=4, 10, 5 | 0 | 0 | 0
  Urea; Increase to Grade 3; n=4, 10, 5 | 0 | 0 | 0
  Urea; Increase to Grade 4; n=4, 10, 5 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Part 2
Description: Blood samples were collected for the analysis of clinical chemistry parameters: glucose, albumin, ALP, ALT, amylase, AST, Dir bil, bilirubin, NT-BNP, calcium, cholesterol, CK, chloride, CO2, creatinine, GGT, HDL and LDL cholesterol, insulin, potassium, LDH, lipase, magnesium, protein, sodium, thyroxine, testosterone, triglycerides (triglyc), troponin I and T, urate and urea. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Participants With CRPC: Participants with Castrate-Resistant Prostate Cancer (CRPC) were administered continuous once daily oral dose of 75 mg GSK525762.
Arm/Group | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Participants
  Glucose; Any grade increase; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Glucose; Any grade increase; n=11,13,23,19,21,12 | 10 | 10 | 20 | 16 | 18 | 9
  Glucose; Increase to Grade 3; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Glucose; Increase to Grade 3; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 1 | 2
  Glucose; Increase to Grade 4; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Glucose; Increase to Grade 4; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin; Any grade increase; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Albumin; Any grade increase; n=11,13,23,19,21,12 | 5 | 6 | 9 | 8 | 7 | 5
  Albumin; Increase to Grade 3; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Albumin; Increase to Grade 3; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 1 | 0
  Albumin; Increase to Grade 4; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Albumin; Increase to Grade 4; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  ALP; Any grade increase; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  ALP; Any grade increase; n=11,13,23,19,21,12 | 3 | 1 | 6 | 3 | 4 | 4
  ALP; Increase to Grade 3; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  ALP; Increase to Grade 3; n=11,13,23,19,21,12 | 0 | 0 | 2 | 0 | 0 | 0
  ALP; Increase to Grade 4; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  ALP; Increase to Grade 4; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  ALT; Any grade increase; n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  ALT; Any grade increase; n=11,14,23,19,21,12 | 3 | 6 | 6 | 5 | 12 | 3
  ALT; Increase to Grade 3; n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  ALT; Increase to Grade 3; n=11,14,23,19,21,12 | 0 | 1 | 0 | 0 | 0 | 0
  ALT; Increase to Grade 4; n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  ALT; Increase to Grade 4; n=11,14,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase; Any grade increase; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Amylase; Any grade increase; n=11,12,22,19,20,12 | 5 | 5 | 9 | 5 | 6 | 1
  Amylase; Increase to Grade 3; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Amylase; Increase to Grade 3; n=11,12,22,19,20,12 | 1 | 2 | 2 | 2 | 2 | 0
  Amylase; Increase to Grade 4; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Amylase; Increase to Grade 4; n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  AST; Any grade increase; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  AST; Any grade increase; n=11,13,23,19,21,12 | 3 | 5 | 10 | 8 | 14 | 6
  AST; Increase to Grade 3; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  AST; Increase to Grade 3; n=11,13,23,19,21,12 | 0 | 0 | 1 | 1 | 3 | 0
  AST; Increase to Grade 4; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  AST; Increase to Grade 4; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Dir bil; Any grade increase; n=11,13,23,19,20,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 20 | 12
  Dir bil; Any grade increase; n=11,13,23,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Dir bil; Increase to Grade 3; n=11,13,23,19,20,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 20 | 12
  Dir bil; Increase to Grade 3; n=11,13,23,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Dir bil; Increase to Grade 4; n=11,13,23,19,20,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 20 | 12
  Dir bil; Increase to Grade 4; n=11,13,23,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin;Any grade increase;n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Bilirubin;Any grade increase;n=11,14,23,19,21,12 | 8 | 10 | 13 | 6 | 13 | 4
  Bilirubin;Increase to Grade 3; n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Bilirubin;Increase to Grade 3; n=11,14,23,19,21,12 | 1 | 1 | 2 | 0 | 3 | 0
  Bilirubin;Increase to Grade 4; n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Bilirubin;Increase to Grade 4; n=11,14,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  NT-BNP; Any grade increase; n=11,12,22,17,15,12: number analyzed (Participants) | 11 | 12 | 22 | 17 | 15 | 12
  NT-BNP; Any grade increase; n=11,12,22,17,15,12 | 0 | 0 | 0 | 0 | 0 | 0
  NT-BNP; Increase to Grade 3; n=11,12,22,17,15,12: number analyzed (Participants) | 11 | 12 | 22 | 17 | 15 | 12
  NT-BNP; Increase to Grade 3; n=11,12,22,17,15,12 | 0 | 0 | 0 | 0 | 0 | 0
  NT-BNP; Increase to Grade 4; n=11,12,22,17,15,12: number analyzed (Participants) | 11 | 12 | 22 | 17 | 15 | 12
  NT-BNP; Increase to Grade 4; n=11,12,22,17,15,12 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Any grade increase; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Calcium; Any grade increase; n=11,13,23,19,21,12 | 6 | 3 | 8 | 4 | 3 | 3
  Calcium; Increase to Grade 3; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Calcium; Increase to Grade 3; n=11,13,23,19,21,12 | 1 | 0 | 2 | 0 | 1 | 0
  Calcium; Increase to Grade 4; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Calcium; Increase to Grade 4; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Cholesterol;Any grade increase;n=10,12,22,19,20,12: number analyzed (Participants) | 10 | 12 | 22 | 19 | 20 | 12
  Cholesterol;Any grade increase;n=10,12,22,19,20,12 | 5 | 2 | 2 | 2 | 9 | 5
  Cholesterol;Increase to Grade3;n=10,12,22,19,20,12: number analyzed (Participants) | 10 | 12 | 22 | 19 | 20 | 12
  Cholesterol;Increase to Grade3;n=10,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Cholesterol;Increase to Grade4;n=10,12,22,19,20,12: number analyzed (Participants) | 10 | 12 | 22 | 19 | 20 | 12
  Cholesterol;Increase to Grade4;n=10,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  CK; Any grade increase; n=9,9,21,17,18,11: number analyzed (Participants) | 9 | 9 | 21 | 17 | 18 | 11
  CK; Any grade increase; n=9,9,21,17,18,11 | 3 | 2 | 4 | 0 | 7 | 5
  CK; Increase to Grade 3; n=9,9,21,17,18,11: number analyzed (Participants) | 9 | 9 | 21 | 17 | 18 | 11
  CK; Increase to Grade 3; n=9,9,21,17,18,11 | 0 | 0 | 0 | 0 | 0 | 0
  CK; Increase to Grade 4; n=9,9,21,17,18,11: number analyzed (Participants) | 9 | 9 | 21 | 17 | 18 | 11
  CK; Increase to Grade 4; n=9,9,21,17,18,11 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride; Any grade increase; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Chloride; Any grade increase; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride; Increase to Grade 3; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Chloride; Increase to Grade 3; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride; Increase to Grade 4; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Chloride; Increase to Grade 4; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  CO2; Any grade increase; n=11,12,23,19,21,12: number analyzed (Participants) | 11 | 12 | 23 | 19 | 21 | 12
  CO2; Any grade increase; n=11,12,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  CO2; Increase to Grade 3; n=11,12,23,19,21,12: number analyzed (Participants) | 11 | 12 | 23 | 19 | 21 | 12
  CO2; Increase to Grade 3; n=11,12,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  CO2; Increase to Grade 4; n=11,12,23,19,21,12: number analyzed (Participants) | 11 | 12 | 23 | 19 | 21 | 12
  CO2; Increase to Grade 4; n=11,12,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine;Any grade increase;n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Creatinine;Any grade increase;n=11,14,23,19,21,12 | 3 | 4 | 9 | 2 | 6 | 3
  Creatinine;Increase to Grade3;n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Creatinine;Increase to Grade3;n=11,14,23,19,21,12 | 0 | 0 | 2 | 0 | 0 | 0
  Creatinine;Increase to Grade4;n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Creatinine;Increase to Grade4;n=11,14,23,19,21,12 | 0 | 0 | 1 | 0 | 0 | 0
  GGT; Any grade increase; n=11,13,22,19,20,12: number analyzed (Participants) | 11 | 13 | 22 | 19 | 20 | 12
  GGT; Any grade increase; n=11,13,22,19,20,12 | 0 | 3 | 7 | 5 | 6 | 1
  GGT; Increase to Grade 3; n=11,13,22,19,20,12: number analyzed (Participants) | 11 | 13 | 22 | 19 | 20 | 12
  GGT; Increase to Grade 3; n=11,13,22,19,20,12 | 0 | 0 | 2 | 2 | 3 | 0
  GGT; Increase to Grade 4; n=11,13,22,19,20,12: number analyzed (Participants) | 11 | 13 | 22 | 19 | 20 | 12
  GGT; Increase to Grade 4; n=11,13,22,19,20,12 | 0 | 0 | 0 | 0 | 1 | 0
  HDL; Any grade increase; n=10,10,22,19,19,12: number analyzed (Participants) | 10 | 10 | 22 | 19 | 19 | 12
  HDL; Any grade increase; n=10,10,22,19,19,12 | 0 | 0 | 0 | 0 | 0 | 0
  HDL; Increase to Grade 3; n=10,10,22,19,19,12: number analyzed (Participants) | 10 | 10 | 22 | 19 | 19 | 12
  HDL; Increase to Grade 3; n=10,10,22,19,19,12 | 0 | 0 | 0 | 0 | 0 | 0
  HDL; Increase to Grade 4;n=10,10,22,19,19,12: number analyzed (Participants) | 10 | 10 | 22 | 19 | 19 | 12
  HDL; Increase to Grade 4;n=10,10,22,19,19,12 | 0 | 0 | 0 | 0 | 0 | 0
  Insulin; Any grade increase; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Insulin; Any grade increase; n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Insulin; Increase to Grade 3; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Insulin; Increase to Grade 3; n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Insulin; Increase to Grade 4; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Insulin; Increase to Grade 4; n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium; Any grade increase; n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Potassium; Any grade increase; n=11,14,23,19,21,12 | 6 | 4 | 10 | 5 | 7 | 7
  Potassium;Increase to Grade3;n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Potassium;Increase to Grade3;n=11,14,23,19,21,12 | 0 | 0 | 1 | 0 | 0 | 1
  Potassium;Increase to Grade4;n=11,14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Potassium;Increase to Grade4;n=11,14,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  LDL; Any grade increase; n=10,10,22,19,19,12: number analyzed (Participants) | 10 | 10 | 22 | 19 | 19 | 12
  LDL; Any grade increase; n=10,10,22,19,19,12 | 0 | 0 | 0 | 0 | 0 | 0
  LDL; Increase to Grade 3; n=10,10,22,19,19,12: number analyzed (Participants) | 10 | 10 | 22 | 19 | 19 | 12
  LDL; Increase to Grade 3; n=10,10,22,19,19,12 | 0 | 0 | 0 | 0 | 0 | 0
  LDL; Increase to Grade 4;n=10,10,22,19,19,12: number analyzed (Participants) | 10 | 10 | 22 | 19 | 19 | 12
  LDL; Increase to Grade 4;n=10,10,22,19,19,12 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase; Any grade increase; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Lipase; Any grade increase; n=11,12,22,19,20,12 | 3 | 5 | 7 | 5 | 4 | 2
  Lipase; Increase to Grade 3;n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Lipase; Increase to Grade 3;n=11,12,22,19,20,12 | 2 | 3 | 0 | 1 | 0 | 0
  Lipase; Increase to Grade 4;n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Lipase; Increase to Grade 4;n=11,12,22,19,20,12 | 0 | 0 | 0 | 1 | 1 | 0
  Magnesium; Any grade increase; n=11,12,22,19,21,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 21 | 12
  Magnesium; Any grade increase; n=11,12,22,19,21,12 | 2 | 2 | 5 | 1 | 4 | 1
  Magnesium; Increase to Grade 3;n=11,12,22,19,21,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 21 | 12
  Magnesium; Increase to Grade 3;n=11,12,22,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Magnesium; Increase to Grade4;n=11,12,22,19,21,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 21 | 12
  Magnesium; Increase to Grade4;n=11,12,22,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Any grade increase; n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Protein; Any grade increase; n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Increase to Grade 3;n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Protein; Increase to Grade 3;n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Protein; Increase to Grade 4;n=11,13,23,19,21,12: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 12
  Protein; Increase to Grade 4;n=11,13,23,19,21,12 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium; Any grade increase; n=11, 14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Sodium; Any grade increase; n=11, 14,23,19,21,12 | 5 | 5 | 8 | 5 | 4 | 5
  Sodium; Increase to Grade 3; n=11, 14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Sodium; Increase to Grade 3; n=11, 14,23,19,21,12 | 0 | 1 | 1 | 2 | 0 | 2
  Sodium; Increase to Grade 4; n=11, 14,23,19,21,12: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 12
  Sodium; Increase to Grade 4; n=11, 14,23,19,21,12 | 1 | 0 | 0 | 0 | 0 | 0
  Thyroxine; Any grade increase;n=7,7,20,15,18,8: number analyzed (Participants) | 7 | 7 | 20 | 15 | 18 | 8
  Thyroxine; Any grade increase;n=7,7,20,15,18,8 | 0 | 0 | 0 | 0 | 0 | 0
  Thyroxine; Increase to Grade3;n=7,7,20,15,18,8: number analyzed (Participants) | 7 | 7 | 20 | 15 | 18 | 8
  Thyroxine; Increase to Grade3;n=7,7,20,15,18,8 | 0 | 0 | 0 | 0 | 0 | 0
  Thyroxine; Increase to Grade4;n=7,7,20,15,18,8: number analyzed (Participants) | 7 | 7 | 20 | 15 | 18 | 8
  Thyroxine; Increase to Grade4;n=7,7,20,15,18,8 | 0 | 0 | 0 | 0 | 0 | 0
  Testosterone; Any grade increase; n=4,3,18,0,1,5: number analyzed (Participants) | 4 | 3 | 18 | 0 | 1 | 5
  Testosterone; Any grade increase; n=4,3,18,0,1,5 | 0 | 0 | 0 | 0 | 0 | 0
  Testosterone; Increase to Grade3; n=4,3,18,0,1,5: number analyzed (Participants) | 4 | 3 | 18 | 0 | 1 | 5
  Testosterone; Increase to Grade3; n=4,3,18,0,1,5 | 0 | 0 | 0 | 0 | 0 | 0
  Testosterone; Increase to Grade4; n=4,3,18,0,1,5: number analyzed (Participants) | 4 | 3 | 18 | 0 | 1 | 5
  Testosterone; Increase to Grade4; n=4,3,18,0,1,5 | 0 | 0 | 0 | 0 | 0 | 0
  Triglyc;Any grade increase;n=10,12,22,19,20,12: number analyzed (Participants) | 10 | 12 | 22 | 19 | 20 | 12
  Triglyc;Any grade increase;n=10,12,22,19,20,12 | 7 | 7 | 15 | 10 | 11 | 8
  Triglyc;Increase to Grade3;n=10,12,22,19,20,12: number analyzed (Participants) | 10 | 12 | 22 | 19 | 20 | 12
  Triglyc;Increase to Grade3;n=10,12,22,19,20,12 | 1 | 0 | 4 | 0 | 1 | 0
  Triglyc;Increase to Grade4;n=10,12,22,19,20,12: number analyzed (Participants) | 10 | 12 | 22 | 19 | 20 | 12
  Triglyc;Increase to Grade4;n=10,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin I; Any grade increase; n=7,6,15,15,14,7: number analyzed (Participants) | 7 | 6 | 15 | 15 | 14 | 7
  Troponin I; Any grade increase; n=7,6,15,15,14,7 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin I; Increase to Grade 3; n=7,6,15,15,14,7: number analyzed (Participants) | 7 | 6 | 15 | 15 | 14 | 7
  Troponin I; Increase to Grade 3; n=7,6,15,15,14,7 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin I; Increase to Grade 4; n=7,6,15,15,14,7: number analyzed (Participants) | 7 | 6 | 15 | 15 | 14 | 7
  Troponin I; Increase to Grade 4; n=7,6,15,15,14,7 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin T;Any grade increase;n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Troponin T;Any grade increase;n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin T;Increase to Grade3;n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Troponin T;Increase to Grade3;n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin T;Increase to Grade4;n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Troponin T;Increase to Grade4;n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Urate; Any grade increase; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Urate; Any grade increase; n=11,12,22,19,20,12 | 0 | 0 | 2 | 0 | 0 | 2
  Urate; Increase to Grade 3; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Urate; Increase to Grade 3; n=11,12,22,19,20,12 | 0 | 0 | 0 | 0 | 0 | 0
  Urate; Increase to Grade 4; n=11,12,22,19,20,12: number analyzed (Participants) | 11 | 12 | 22 | 19 | 20 | 12
  Urate; Increase to Grade 4; n=11,12,22,19,20,12 | 0 | 0 | 2 | 0 | 0 | 2
  Urea; Any grade increase; n=11,14,23,17,17,11: number analyzed (Participants) | 11 | 14 | 23 | 17 | 17 | 11
  Urea; Any grade increase; n=11,14,23,17,17,11 | 0 | 0 | 0 | 0 | 0 | 0
  Urea; Increase to Grade 3; n=11,14,23,17,17,11: number analyzed (Participants) | 11 | 14 | 23 | 17 | 17 | 11
  Urea; Increase to Grade 3; n=11,14,23,17,17,11 | 0 | 0 | 0 | 0 | 0 | 0
  Urea; Increase to Grade 4;n=11,14,23,17,17,11: number analyzed (Participants) | 11 | 14 | 23 | 17 | 17 | 11
  Urea; Increase to Grade 4;n=11,14,23,17,17,11 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Besylate Sub-study
Description: Blood samples were collected for the analysis of clinical chemistry parameters: glucose, albumin, ALP, ALT, amylase, AST, Dir bil, bilirubin, NT-BNP, calcium, cholesterol, CK, chloride, CO2, creatinine, GGT, HDL and LDL cholesterol, insulin, potassium, LDH, lipase, magnesium, protein, sodium, thyroxine, testosterone, triglycerides, troponin I and T, urate and urea. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.87 months of drug exposure
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  Glucose; Any grade increase; n=5,5 | 4 | 5
  Glucose; Increase to Grade 3; n=5,5 | 0 | 0
  Glucose; Increase to Grade 4; n=5,5 | 0 | 0
  Albumin; Any grade increase; n=5,5 | 3 | 3
  Albumin; Increase to Grade 3; n=5,5 | 1 | 0
  Albumin; Increase to Grade 4; n=5,5 | 0 | 0
  ALP; Any grade increase; n=5,5 | 1 | 0
  ALP; Increase to Grade 3; n=5,5 | 0 | 0
  ALP; Increase to Grade 4; n=5,5 | 0 | 0
  ALT; Any grade increase; n=5,5 | 1 | 1
  ALT; Increase to Grade 3; n=5,5 | 0 | 0
  ALT; Increase to Grade 4; n=5,5 | 0 | 0
  Amylase; Any grade increase; n=5,5 | 0 | 0
  Amylase; Increase to Grade 3; n=5,5 | 0 | 0
  Amylase; Increase to Grade 4; n=5,5 | 0 | 0
  AST; Any grade increase; n=5,5 | 2 | 1
  AST; Increase to Grade 3; n=5,5 | 0 | 0
  AST; Increase to Grade 4; n=5,5 | 0 | 0
  Dir bil; Any grade increase; n=5,5 | 0 | 0
  Dir bil; Increase to Grade 3; n=5,5 | 0 | 0
  Dir bil; Increase to Grade 4; n=5,5 | 0 | 0
  Bilirubin; Any grade increase; n=5,5 | 3 | 4
  Bilirubin; Increase to Grade 3; n=5,5 | 1 | 2
  Bilirubin; Increase to Grade 4; n=5,5 | 0 | 0
  NT-BNP; Any grade increase; n=5,5 | 0 | 0
  NT-BNP; Increase to Grade 3; n=5,5 | 0 | 0
  NT-BNP; Increase to Grade 4; n=5,5 | 0 | 0
  Calcium; Any grade increase; n=5,5 | 1 | 2
  Calcium; Increase to Grade 3; n=5,5 | 0 | 0
  Calcium; Increase to Grade 4; n=5,5 | 0 | 0
  Cholesterol; Any grade increase; n=5,3: number analyzed (Participants) | 5 | 3
  Cholesterol; Any grade increase; n=5,3 | 1 | 0
  Cholesterol; Increase to Grade 3; n=5,3: number analyzed (Participants) | 5 | 3
  Cholesterol; Increase to Grade 3; n=5,3 | 0 | 0
  Cholesterol; Increase to Grade 4; n=5,3: number analyzed (Participants) | 5 | 3
  Cholesterol; Increase to Grade 4; n=5,3 | 0 | 0
  CK; Any grade increase; n=5,5 | 2 | 0
  CK; Increase to Grade 3; n=5,5 | 0 | 0
  CK; Increase to Grade 4; n=5,5 | 0 | 0
  Chloride; Any grade increase; n=5,5 | 0 | 0
  Chloride; Increase to Grade 3; n=5,5 | 0 | 0
  Chloride; Increase to Grade 4; n=5,5 | 0 | 0
  CO2; Any grade increase; n=5,5 | 0 | 0
  CO2; Increase to Grade 3; n=5,5 | 0 | 0
  CO2; Increase to Grade 4; n=5,5 | 0 | 0
  Creatinine; Any grade increase; n=5,5 | 1 | 1
  Creatinine; Increase to Grade 3; n=5,5 | 0 | 0
  Creatinine; Increase to Grade 4; n=5,5 | 0 | 0
  GGT; Any grade increase; n=5,5 | 0 | 0
  GGT; Increase to Grade 3; n=5,5 | 0 | 0
  GGT; Increase to Grade 4; n=5,5 | 0 | 0
  HDL; Any grade increase; n=5,3: number analyzed (Participants) | 5 | 3
  HDL; Any grade increase; n=5,3 | 0 | 0
  HDL; Increase to Grade 3; n=5,3: number analyzed (Participants) | 5 | 3
  HDL; Increase to Grade 3; n=5,3 | 0 | 0
  HDL; Increase to Grade 4; n=5,3: number analyzed (Participants) | 5 | 3
  HDL; Increase to Grade 4; n=5,3 | 0 | 0
  Insulin; Any grade increase; n=5,5 | 0 | 0
  Insulin; Increase to Grade 3; n=5,5 | 0 | 0
  Insulin; Increase to Grade 4; n=5,5 | 0 | 0
  Potassium; Any grade increase; n=5,5 | 3 | 3
  Potassium; Increase to Grade 3; n=5,5 | 0 | 0
  Potassium; Increase to Grade 4; n=5,5 | 0 | 0
  LDL; Any grade increase; n=5,3: number analyzed (Participants) | 5 | 3
  LDL; Any grade increase; n=5,3 | 0 | 0
  LDL; Increase to Grade 3; n=5,3: number analyzed (Participants) | 5 | 3
  LDL; Increase to Grade 3; n=5,3 | 0 | 0
  LDL; Increase to Grade 4; n=5,3: number analyzed (Participants) | 5 | 3
  LDL; Increase to Grade 4; n=5,3 | 0 | 0
  Lipase; Any grade increase; n=5,4: number analyzed (Participants) | 5 | 4
  Lipase; Any grade increase; n=5,4 | 0 | 0
  Lipase; Increase to Grade 3; n=5,4: number analyzed (Participants) | 5 | 4
  Lipase; Increase to Grade 3; n=5,4 | 0 | 0
  Lipase; Increase to Grade 4;n=5,4: number analyzed (Participants) | 5 | 4
  Lipase; Increase to Grade 4;n=5,4 | 0 | 0
  Magnesium; Any grade increase; n=5,5 | 2 | 1
  Magnesium; Increase to Grade 3; n=5,5 | 0 | 1
  Magnesium; Increase to Grade 4; n=5,5 | 0 | 0
  Protein; Any grade increase; n=5,5 | 0 | 0
  Protein; Increase to Grade 3; n=5,5 | 0 | 0
  Protein; Increase to Grade 4; n=5,5 | 0 | 0
  Sodium; Any grade increase; n=5,5 | 2 | 3
  Sodium; Increase to Grade 3; n=5,5 | 0 | 1
  Sodium; Increase to Grade 4; n=5,5 | 0 | 0
  Thyroxine; Any grade increase; n=5,3: number analyzed (Participants) | 5 | 3
  Thyroxine; Any grade increase; n=5,3 | 0 | 0
  Thyroxine; Increase to Grade 3; n=5,3: number analyzed (Participants) | 5 | 3
  Thyroxine; Increase to Grade 3; n=5,3 | 0 | 0
  Thyroxine; Increase to Grade 4; n=5,3: number analyzed (Participants) | 5 | 3
  Thyroxine; Increase to Grade 4; n=5,3 | 0 | 0
  Testosterone; Any grade increase; n=2,1: number analyzed (Participants) | 2 | 1
  Testosterone; Any grade increase; n=2,1 | 0 | 0
  Testosterone; Increase to Grade 3; n=2,1: number analyzed (Participants) | 2 | 1
  Testosterone; Increase to Grade 3; n=2,1 | 0 | 0
  Testosterone; Increase to Grade 4; n=2,1: number analyzed (Participants) | 2 | 1
  Testosterone; Increase to Grade 4; n=2,1 | 0 | 0
  Triglycerides; Any grade increase; n=5,3: number analyzed (Participants) | 5 | 3
  Triglycerides; Any grade increase; n=5,3 | 1 | 2
  Triglycerides; Increase to Grade 3; n=5,3: number analyzed (Participants) | 5 | 3
  Triglycerides; Increase to Grade 3; n=5,3 | 0 | 0
  Triglycerides; Increase to Grade 4; n=5,3: number analyzed (Participants) | 5 | 3
  Triglycerides; Increase to Grade 4; n=5,3 | 0 | 0
  Troponin I; Any grade increase; n=1,0: number analyzed (Participants) | 1 | 0
  Troponin I; Any grade increase; n=1,0 | 0 |
  Troponin I; Increase to Grade 3; n=1,0: number analyzed (Participants) | 1 | 0
  Troponin I; Increase to Grade 3; n=1,0 | 0 |
  Troponin I; Increase to Grade 4; n=1,0: number analyzed (Participants) | 1 | 0
  Troponin I; Increase to Grade 4; n=1,0 | 0 |
  Troponin T; Any grade increase; n=5,5 | 0 | 0
  Troponin T; Increase to Grade 3; n=5,5 | 0 | 0
  Troponin T; Increase to Grade 4; n=5,5 | 0 | 0
  Urate; Any grade increase; n=5,5 | 0 | 0
  Urate; Increase to Grade 3; n=5,5 | 0 | 0
  Urate; Increase to Grade 4; n=5,5 | 0 | 0
  Urea; Any grade increase; n=5,5 | 0 | 0
  Urea; Increase to Grade 3; n=5,5 | 0 | 0
  Urea; Increase to Grade 4; n=5,5 | 0 | 0

16. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Part 1 QD
Description: Blood samples were collected for the analysis of hematology parameters: activated partial thromboplastin time (aPTT), platelet count, red blood cell count (RBC), white blood cell count (WBC), prothrombin international normalized ratio (INR), prothrombin time (PT), fibrinogen (Fib), hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.38 months of drug exposure
Population: All Treated Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 2 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants
  Basophils;Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils;Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils;Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils;Increase to Grade3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin;Any grade increase | 1 | 1 | 0 | 2 | 2 | 2 | 21 | 7
  Hemoglobin;Increase to Grade 3; n=2,4,1,3,4,9,32,9 | 0 | 0 | 0 | 0 | 1 | 1 | 9 | 1
  Hemoglobin;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  INR; Any grade increase | 2 | 2 | 1 | 0 | 0 | 1 | 21 | 2
  INR;Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  INR; Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes;Any grade increase | 1 | 2 | 1 | 0 | 2 | 5 | 19 | 4
  Lymphocytes;Increase to Grade3 | 0 | 1 | 0 | 0 | 0 | 2 | 8 | 1
  Lymphocytes;Increase to Grade4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Monocytes;Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes;Increase to Grade3 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 0
  Monocytes;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils;Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  Neutrophils;Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophils;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets;Any grade increase | 0 | 1 | 0 | 0 | 2 | 5 | 26 | 8
  Platelets;Increase to Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 11 | 5
  Platelets;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2
  PT; Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PT; Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PT; Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC; Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC;Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC; Any grade increase | 0 | 1 | 0 | 0 | 0 | 3 | 11 | 5
  WBC; Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  WBC; Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Fib; Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
  Fib;Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fib;Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  aPTT; Any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 2
  aPTT; Increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  aPTT; Increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Part 1 BID
Description: Blood samples were collected for the analysis of hematology parameters: aPTT, platelet count, RBC, WBC, INR, PT, Fib, hemoglobin, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: GSK525762 40 mg BID: Participants were administered once daily oral dose of 40 mg GSK525762.
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  Basophils; Any grade increase; n=4,10,5 | 0 | 0 | 0
  Basophils; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  Basophils; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  Eosinophils; Any grade increase; n=4,10,5 | 0 | 0 | 0
  Eosinophils; Increase to Grade3; n=4,10,5 | 0 | 0 | 0
  Eosinophils; Increase to Grade4; n=4,10,5 | 0 | 0 | 0
  Hemoglobin; Any grade increase; n=4,10,5 | 4 | 8 | 4
  Hemoglobin; Increase to Grade 3; n=4,10,5 | 0 | 3 | 2
  Hemoglobin; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  INR; Any grade increase; n=4,10,5 | 0 | 6 | 3
  INR; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  INR; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  Lymphocytes; Any grade increase; n=4,10,5 | 2 | 8 | 2
  Lymphocytes; Increase to Grade3; n=4,10,5 | 0 | 4 | 0
  Lymphocytes; Increase to Grade4; n=4,10,5 | 0 | 0 | 0
  Monocytes; Any grade increase; n=4,10,5 | 0 | 0 | 0
  Monocytes;Increase to Grade3; n=4,10,5 | 0 | 0 | 0
  Monocytes; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  Neutrophils; Any grade increase; n=4,10,5 | 0 | 0 | 1
  Neutrophils; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  Neutrophils; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  Platelets; Any grade increase; n=4,10,5 | 1 | 10 | 5
  Platelets; Increase to Grade 3; n=4,10,5 | 0 | 2 | 2
  Platelets; Increase to Grade 4; n=4,10,5 | 0 | 0 | 1
  PT; Any grade increase;n=4,10,5 | 0 | 0 | 0
  PT; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  PT; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  RBC; Any grade increase; n=4,10,5 | 0 | 0 | 0
  RBC; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  RBC; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  WBC; Any grade increase; n=4,10,5 | 1 | 0 | 1
  WBC; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  WBC; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  Fib; Any grade increase; n=4,10,5 | 0 | 0 | 0
  Fib; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  Fib; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0
  aPTT; Any grade increase; n=4,10,5 | 0 | 5 | 2
  aPTT; Increase to Grade 3; n=4,10,5 | 0 | 0 | 0
  aPTT; Increase to Grade 4; n=4,10,5 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Part 2
Description: as for outcome 17
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Participants
  Basophils; Any grade increase; n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Basophils; Any grade increase; n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils; Increase to Grade3; n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Basophils; Increase to Grade3; n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils; Increase to Grade4; n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Basophils; Increase to Grade4; n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils;Any grade increase;n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Eosinophils;Any grade increase;n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils;Increase to Grade3;n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Eosinophils;Increase to Grade3;n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils;Increase to Grade4;n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Eosinophils;Increase to Grade4;n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin;Any grade increase;n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Hemoglobin;Any grade increase;n=11,14,23,19,21,13 | 6 | 10 | 18 | 10 | 18 | 6
  Hemoglobin;Increase to Grade3;n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Hemoglobin;Increase to Grade3;n=11,14,23,19,21,13 | 3 | 2 | 9 | 4 | 5 | 3
  Hemoglobin;Increase to Grade4;n=11,14, 23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Hemoglobin;Increase to Grade4;n=11,14, 23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  INR; Any grade increase; n=11,12,21,17,18,12: number analyzed (Participants) | 11 | 12 | 21 | 17 | 18 | 12
  INR; Any grade increase; n=11,12,21,17,18,12 | 8 | 6 | 13 | 8 | 11 | 7
  INR; Increase to Grade3; n=11,12,21,17,18,12: number analyzed (Participants) | 11 | 12 | 21 | 17 | 18 | 12
  INR; Increase to Grade3; n=11,12,21,17,18,12 | 0 | 0 | 0 | 0 | 0 | 0
  INR; Increase to Grade4; n=11,12,21,17,18,12: number analyzed (Participants) | 11 | 12 | 21 | 17 | 18 | 12
  INR; Increase to Grade4; n=11,12,21,17,18,12 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes;Any grade increase;n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Lymphocytes;Any grade increase;n=11,13,23,19,21,13 | 8 | 7 | 14 | 9 | 13 | 6
  Lymphocytes;Increase to Grade3;n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Lymphocytes;Increase to Grade3;n=11,13,23,19,21,13 | 2 | 2 | 6 | 2 | 1 | 0
  Lymphocytes;Increase to Grade4;n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Lymphocytes;Increase to Grade4;n=11,13,23,19,21,13 | 0 | 1 | 0 | 0 | 0 | 0
  Monocytes; Any grade increase; n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Monocytes; Any grade increase; n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes;Increase to Grade3; n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Monocytes;Increase to Grade3; n=11,13,23,19,21,13 | 0 | 0 | 00 | 0 | 0 | 0
  Monocytes; Increase to Grade4; n=11,13,23,19,21,13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  Monocytes; Increase to Grade4; n=11,13,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils;Any grade increase;n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Neutrophils;Any grade increase;n=11,14,23,19,21,13 | 4 | 4 | 8 | 3 | 6 | 1
  Neutrophils;Increase to Grade3;n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Neutrophils;Increase to Grade3;n=11,14,23,19,21,13 | 1 | 1 | 0 | 2 | 1 | 0
  Neutrophils;Increase to Grade4;n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Neutrophils;Increase to Grade4;n=11,14,23,19,21,13 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets; Any grade increase; n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Platelets; Any grade increase; n=11,14,23,19,21,13 | 7 | 12 | 20 | 17 | 18 | 7
  Platelets; Increase to Grade3; n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Platelets; Increase to Grade3; n=11,14,23,19,21,13 | 4 | 4 | 5 | 6 | 6 | 0
  Platelets; Increase to Grade4; n=11,14,23,19,21,13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  Platelets; Increase to Grade4; n=11,14,23,19,21,13 | 2 | 3 | 8 | 4 | 2 | 0
  PT; Any grade increase;n=10,10, 18, 17, 18, 12: number analyzed (Participants) | 10 | 10 | 18 | 17 | 18 | 12
  PT; Any grade increase;n=10,10, 18, 17, 18, 12 | 0 | 0 | 0 | 0 | 0 | 0
  PT; Increase to Grade 3; n=10,10, 18, 17, 18, 12: number analyzed (Participants) | 10 | 10 | 18 | 17 | 18 | 12
  PT; Increase to Grade 3; n=10,10, 18, 17, 18, 12 | 0 | 0 | 0 | 0 | 0 | 0
  PT; Increase to Grade 4; n=10,10, 18, 17, 18, 12: number analyzed (Participants) | 10 | 10 | 18 | 17 | 18 | 12
  PT; Increase to Grade 4; n=10,10, 18, 17, 18, 12 | 0 | 0 | 0 | 0 | 0 | 0
  RBC; Any grade increase; n=11, 13, 23, 19, 21, 13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  RBC; Any grade increase; n=11, 13, 23, 19, 21, 13 | 0 | 0 | 0 | 0 | 0 | 0
  RBC; Increase to Grade 3; n=11, 13, 23, 19, 21, 13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  RBC; Increase to Grade 3; n=11, 13, 23, 19, 21, 13 | 0 | 0 | 0 | 0 | 0 | 0
  RBC; Increase to Grade 4; n=11, 13, 23, 19, 21, 13: number analyzed (Participants) | 11 | 13 | 23 | 19 | 21 | 13
  RBC; Increase to Grade 4; n=11, 13, 23, 19, 21, 13 | 0 | 0 | 0 | 0 | 0 | 0
  WBC; Any grade increase; n=11, 14, 23, 19, 21, 13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  WBC; Any grade increase; n=11, 14, 23, 19, 21, 13 | 7 | 5 | 9 | 5 | 6 | 3
  WBC; Increase to Grade 3; n=11, 14, 23, 19, 21, 13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  WBC; Increase to Grade 3; n=11, 14, 23, 19, 21, 13 | 1 | 0 | 1 | 1 | 0 | 0
  WBC; Increase to Grade 4; n=11, 14, 23, 19, 21, 13: number analyzed (Participants) | 11 | 14 | 23 | 19 | 21 | 13
  WBC; Increase to Grade 4; n=11, 14, 23, 19, 21, 13 | 0 | 0 | 0 | 0 | 0 | 0
  Fib; Any grade increase; n=11, 11, 21, 17, 18, 12: number analyzed (Participants) | 11 | 11 | 21 | 17 | 18 | 12
  Fib; Any grade increase; n=11, 11, 21, 17, 18, 12 | 2 | 0 | 1 | 0 | 0 | 1
  Fib; Increase to Grade 3; n=11, 11, 21, 17, 18, 12: number analyzed (Participants) | 11 | 11 | 21 | 17 | 18 | 12
  Fib; Increase to Grade 3; n=11, 11, 21, 17, 18, 12 | 1 | 0 | 0 | 0 | 0 | 0
  Fib; Increase to Grade 4; n=11, 11, 21, 17, 18, 12: number analyzed (Participants) | 11 | 11 | 21 | 17 | 18 | 12
  Fib; Increase to Grade 4; n=11, 11, 21, 17, 18, 12 | 0 | 0 | 0 | 0 | 0 | 0
  aPTT; Any grade increase; n=11,12,21,17,18,12: number analyzed (Participants) | 11 | 12 | 21 | 17 | 18 | 12
  aPTT; Any grade increase; n=11,12,21,17,18,12 | 4 | 4 | 1 | 3 | 5 | 4
  aPTT; Increase to Grade3; n=11,12,21, 17, 18, 12: number analyzed (Participants) | 11 | 12 | 21 | 17 | 18 | 12
  aPTT; Increase to Grade3; n=11,12,21, 17, 18, 12 | 0 | 0 | 0 | 1 | 0 | 0
  aPTT; Increase to Grade4; n=11,12,21,17,18,12: number analyzed (Participants) | 11 | 12 | 21 | 17 | 18 | 12
  aPTT; Increase to Grade4; n=11,12,21,17,18,12 | 0 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Besylate Sub-study
Description: as for outcome 17
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  Basophils; Any grade increase | 0 | 0
  Basophils; Increase to Grade 3 | 0 | 0
  Basophils; Increase to Grade 4 | 0 | 0
  Eosinophils; Any grade increase | 0 | 0
  Eosinophils; Increase to Grade 3 | 0 | 0
  Eosinophils; Increase to Grade 4 | 0 | 0
  Hemoglobin; Any grade increase | 4 | 3
  Hemoglobin; Increase to Grade 3 | 2 | 2
  Hemoglobin; Increase to Grade 4 | 0 | 0
  INR; Any grade increase | 1 | 1
  INR; Increase to Grade 3 | 0 | 0
  INR; Increase to Grade 4 | 0 | 0
  Lymphocytes; Any grade increase | 3 | 4
  Lymphocytes; Increase to Grade 3 | 1 | 0
  Lymphocytes; Increase to Grade 4 | 2 | 0
  Monocytes; Any grade increase | 0 | 0
  Monocytes; Increase to Grade 3 | 0 | 0
  Monocytes; Increase to Grade 4 | 0 | 0
  Neutrophils; Any grade increase | 1 | 1
  Neutrophils; Increase to Grade 3 | 0 | 0
  Neutrophils; Increase to Grade 4 | 0 | 0
  Platelets; Any grade increase | 5 | 5
  Platelets; Increase to Grade 3 | 0 | 2
  Platelets; Increase to Grade 4 | 3 | 1
  PT; Any grade increase | 0 | 0
  PT; Increase to Grade 3 | 0 | 0
  PT; Increase to Grade 4 | 0 | 0
  RBC; Any grade increase | 0 | 0
  RBC; Increase to Grade 3 | 0 | 0
  RBC; Increase to Grade 4 | 0 | 0
  WBC; Any grade increase | 3 | 1
  WBC; Increase to Grade 3 | 0 | 0
  WBC; Increase to Grade 4 | 0 | 0
  Fib; Any grade increase | 0 | 0
  Fib; Increase to Grade 3 | 0 | 0
  Fib; Increase to Grade 4 | 0 | 0
  aPTT; Any grade increase | 4 | 2
  aPTT; Increase to Grade 3 | 0 | 0
  aPTT; Increase to Grade 4 | 0 | 0

20. Primary Outcome: Number of Participants With Maximum Urinalysis Change From Baseline-Part 1 QD
Description: Urine samples were collected for the analysis of following urine parameters: potential of hydrogen (pH), glucose, protein, occult blood, ketones, specific gravity, erythrocytes and leukocytes. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Only parameters and time points with non-zero values for any increase have been presented.
Time Frame: Baseline (pre-dose Week1 Day1) and Weeks 5, 9, 17, 25, 33, 41, 49 and discharge/progression (disc/prog)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants
  Cellular casts; Week 9; n=0,0, 0, 0, 0,1,4,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1
  Cellular casts; Week 9; n=0,0, 0, 0, 0,1,4,1 |  |  |  |  |  | 0 | 1 | 1
  Cellular casts; Week 17; n=0,0, 0, 0, 0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cellular casts; Week 17; n=0,0, 0, 0, 0,0,1,0 |  |  |  |  |  |  | 1 |
  Cellular casts; Disc/Prog; n=0,0,0,0,0,1,5,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1
  Cellular casts; Disc/Prog; n=0,0,0,0,0,1,5,1 |  |  |  |  |  | 0 | 1 | 0
  Hyaline casts;Week 5; n=0,1,0,0,1,2,5,3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 2 | 5 | 3
  Hyaline casts;Week 5; n=0,1,0,0,1,2,5,3 |  | 0 |  |  | 0 | 0 | 2 | 1
  Hyaline casts;Week 9; n=0,1,0, 0,0,1,5,3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 3
  Hyaline casts;Week 9; n=0,1,0, 0,0,1,5,3 |  | 0 |  |  |  | 0 | 0 | 1
  Glucose;Week 5; n=1,2,1,3,2,7,20,7: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 7 | 20 | 7
  Glucose;Week 5; n=1,2,1,3,2,7,20,7 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Glucose;Week 9; n=1, 1, 0, 1,1,3,12,5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 3 | 12 | 5
  Glucose;Week 9; n=1, 1, 0, 1,1,3,12,5 | 0 | 0 |  | 0 | 0 | 0 | 1 | 1
  Glucose;Week 25; n=0,1,0,0,0,0,3,1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
  Glucose;Week 25; n=0,1,0,0,0,0,3,1 |  | 0 |  |  |  |  | 0 | 1
  Glucose;Disc/Prog; n=0, 1, 0,1,0,3,17,2: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 3 | 17 | 2
  Glucose;Disc/Prog; n=0, 1, 0,1,0,3,17,2 | 0 | 0 | 0 | 1 |  | 0 | 1 | 0
  Ketones;Week 5; n=1,2,1,3,2,7,20,7: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 7 | 20 | 7
  Ketones;Week 5; n=1,2,1,3,2,7,20,7 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Ketones;Week 9; n=1,1,0,1,1,3,12,5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 3 | 12 | 5
  Ketones;Week 9; n=1,1,0,1,1,3,12,5 | 0 | 0 |  | 0 | 0 | 0 | 2 | 0
  Occult blood;Week 5; n=1,2,1,3,2,7,17,7: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 7 | 17 | 7
  Occult blood;Week 5; n=1,2,1,3,2,7,17,7 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  Occult blood;Week 9; n=1,1,0,1,1,3,11,5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 3 | 11 | 5
  Occult blood;Week 9; n=1,1,0,1,1,3,11,5 | 0 | 0 |  | 0 | 0 | 0 | 3 | 0
  Occult blood;Week 17; n=0, 1,0,0,0,0,5,3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 3
  Occult blood;Week 17; n=0, 1,0,0,0,0,5,3 |  | 0 |  |  |  |  | 1 | 0
  Occult blood;Week 25; n=0,1,0,0,0,0,3,1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
  Occult blood;Week 25; n=0,1,0,0,0,0,3,1 |  | 0 |  |  |  |  | 1 | 0
  Occult blood;Week 33; n=0,1,0,0,0,0,2,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Occult blood;Week 33; n=0,1,0,0,0,0,2,0 |  | 0 |  |  |  |  | 1 |
  Occult blood;Disc/Prog; n=0,1,0,1,0,3,17,2: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 3 | 17 | 2
  Occult blood;Disc/Prog; n=0,1,0,1,0,3,17,2 |  | 0 |  | 0 |  | 0 | 2 | 0
  pH;Week 5; n=1, 2, 1, 3,2,7,20,7: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 7 | 20 | 7
  pH;Week 5; n=1, 2, 1, 3,2,7,20,7 | 0 | 0 | 0 | 1 | 0 | 5 | 6 | 3
  pH;Week 9; n=1,1,0,1,1,3,12,5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 3 | 12 | 5
  pH;Week 9; n=1,1,0,1,1,3,12,5 | 0 | 1 | 0 | 1 | 0 | 2 | 8 | 2
  pH;Week 25; n=0,1,0,0,0,0,3,1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
  pH;Week 25; n=0,1,0,0,0,0,3,1 | 0 | 1 | 0 | 0 |  |  | 1 | 1
  pH;Week 33; n=0,1,0,0,0,0,2,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  pH;Week 33; n=0,1,0,0,0,0,2,0 |  | 1 |  |  |  |  | 0 |
  pH;Disc/Prog; n=0,1,0,1,0,3,17,2: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 3 | 17 | 2
  pH;Disc/Prog; n=0,1,0,1,0,3,17,2 |  | 1 |  | 0 |  | 1 | 9 | 1
  Protein;Week 5; n=1, 2,1,3,2,7,20,7: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 7 | 20 | 7
  Protein;Week 5; n=1, 2,1,3,2,7,20,7 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 4
  Protein;Week 9; n=1,1,0,1,1,3,12,5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 3 | 12 | 5
  Protein;Week 9; n=1,1,0,1,1,3,12,5 | 0 | 1 |  | 0 | 0 | 1 | 7 | 3
  Protein;Week 17; n=0,1,0,0,0,0,5,3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 3
  Protein;Week 17; n=0,1,0,0,0,0,5,3 |  | 0 |  |  |  |  | 1 | 0
  Protein;Week 25; n=0,1,0,0,0,0,3,1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
  Protein;Week 25; n=0,1,0,0,0,0,3,1 |  | 0 |  |  |  |  | 1 | 0
  Protein;Disc/Prog; n=0,1,0,1,0,3,17,2: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 3 | 17 | 2
  Protein;Disc/Prog; n=0,1,0,1,0,3,17,2 |  | 0 |  | 0 |  | 0 | 5 | 1
  Specific gravity;Week 5; n=1,2,1,3,2,7,20,7: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 7 | 20 | 7
  Specific gravity;Week 5; n=1,2,1,3,2,7,20,7 | 1 | 1 | 0 | 2 | 2 | 5 | 7 | 5
  Specific gravity;Week 9; n=1,1,0,1,1,3,12,5: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 3 | 12 | 5
  Specific gravity;Week 9; n=1,1,0,1,1,3,12,5 | 1 | 0 |  | 0 | 0 | 2 | 6 | 4
  Specific gravity;Week 17; n=0,1,0,0,0,0,5,3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 3
  Specific gravity;Week 17; n=0,1,0,0,0,0,5,3 |  | 1 |  |  |  |  | 4 | 2
  Specific gravity;Week 25; n=0,1,0,0,0,0,3,1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
  Specific gravity;Week 25; n=0,1,0,0,0,0,3,1 |  | 1 |  |  |  |  | 1 | 0
  Specific gravity;Week 33; n=0,1,0,0,0,0,2,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Specific gravity;Week 33; n=0,1,0,0,0,0,2,0 |  | 1 |  |  |  |  | 1 |
  Specific gravity;Disc/Prog; n=0,1,0,1,0,3,16,2: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 3 | 16 | 2
  Specific gravity;Disc/Prog; n=0,1,0,1,0,3,16,2 |  | 1 |  | 1 |  | 1 | 6 | 1
  Specific gravity;Week 41; n=0,0,0,0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Specific gravity;Week 41; n=0,0,0,0,0,0,1,0 |  |  |  |  |  |  | 1 |
  Specific gravity;Week 49; n=0,0,0,0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Specific gravity;Week 49; n=0,0,0,0,0,0,1,0 |  |  |  |  |  |  | 1 |
  Leukocytes;Week 5; n=1,2,1,2,2,6,11,6: number analyzed (Participants) | 1 | 2 | 1 | 2 | 2 | 6 | 11 | 6
  Leukocytes;Week 5; n=1,2,1,2,2,6,11,6 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 2
  Leukocytes;Week 9; n=1,1,0,1,1,1,6,4: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 1 | 6 | 4
  Leukocytes;Week 9; n=1,1,0,1,1,1,6,4 | 0 | 0 |  | 0 | 1 | 0 | 3 | 1
  Leukocytes;Week 17; n=0,1,0,0,0,0,1,2: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Leukocytes;Week 17; n=0,1,0,0,0,0,1,2 |  | 0 |  |  |  |  | 1 | 0
  Leukocytes;Disc/Prog; n=0,1,0,1,0,2,6,1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 6 | 1
  Leukocytes;Disc/Prog; n=0,1,0,1,0,2,6,1 |  | 0 |  | 0 |  | 0 | 4 | 1

21. Primary Outcome: Number of Participants With Maximum Urinalysis Change From Baseline Data-Part 1 BID
Description: Urine samples were collected for the analysis of following urine parameters: pH, glucose, protein, occult blood, ketones, specific gravity, erythrocytes and leukocytes. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Only parameters and time points with non-zero values for any increase have been presented.
Time Frame: Baseline (pre-dose Week1 Day1) and Weeks 5,9,17 and discharge/progression
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  Glucose; Week 5;n=2,7,3: number analyzed (Participants) | 2 | 7 | 3
  Glucose; Week 5;n=2,7,3 | 0 | 0 | 1
  Glucose; Week 9;n=0,4,2: number analyzed (Participants) | 0 | 4 | 2
  Glucose; Week 9;n=0,4,2 |  | 1 | 0
  Glucose; Week 17;n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Glucose; Week 17;n=0,2,0 |  | 1 |
  Glucose; disc/prog;n=0,6,1: number analyzed (Participants) | 0 | 6 | 1
  Glucose; disc/prog;n=0,6,1 |  | 1 | 0
  Ketones; Week 5;n=2,7,3: number analyzed (Participants) | 2 | 7 | 3
  Ketones; Week 5;n=2,7,3 | 0 | 1 | 0
  Ketones; Week 17;n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Ketones; Week 17;n=0,2,0 |  | 1 |
  Occult blood; Week 5;n=2,7,3: number analyzed (Participants) | 2 | 7 | 3
  Occult blood; Week 5;n=2,7,3 | 0 | 2 | 0
  Occult blood; Week 9;n=0,4,2: number analyzed (Participants) | 0 | 4 | 2
  Occult blood; Week 9;n=0,4,2 |  | 1 | 0
  Occult blood; disc/prog;n=0,6,1: number analyzed (Participants) | 0 | 6 | 1
  Occult blood; disc/prog;n=0,6,1 |  | 2 | 0
  pH; Week 5;n=2,7,3: number analyzed (Participants) | 2 | 7 | 3
  pH; Week 5;n=2,7,3 | 2 | 4 | 2
  pH; Week 9;n=0,4,2: number analyzed (Participants) | 0 | 4 | 2
  pH; Week 9;n=0,4,2 |  | 4 | 1
  pH; Week 17;n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  pH; Week 17;n=0,2,0 |  | 1 |
  pH; disc/prog;n=0,7,1: number analyzed (Participants) | 0 | 7 | 1
  pH; disc/prog;n=0,7,1 |  | 4 | 1
  Protein; Week 5;n=2,7,3: number analyzed (Participants) | 2 | 7 | 3
  Protein; Week 5;n=2,7,3 | 0 | 3 | 1
  Protein; Week 9;n=0,4,2: number analyzed (Participants) | 0 | 4 | 2
  Protein; Week 9;n=0,4,2 |  | 2 | 0
  Protein; Week 17;n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Protein; Week 17;n=0,2,0 |  | 2 |
  Protein; disc/prog;n=0,7,1: number analyzed (Participants) | 0 | 7 | 1
  Protein; disc/prog;n=0,7,1 |  | 1 | 1
  Erythrocytes; Week 5;n=1,5,1: number analyzed (Participants) | 1 | 5 | 1
  Erythrocytes; Week 5;n=1,5,1 | 1 | 4 | 1
  Erythrocytes; Week 9;n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  Erythrocytes; Week 9;n=0,1,1 |  | 0 | 1
  Erythrocytes; Week 17;n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Erythrocytes; Week 17;n=0,1,0 |  | 1 |
  Specific gravity; Week 5;n=2,7,3: number analyzed (Participants) | 2 | 7 | 3
  Specific gravity; Week 5;n=2,7,3 | 2 | 1 | 2
  Specific gravity; Week 9;n=0,4,2: number analyzed (Participants) | 0 | 4 | 2
  Specific gravity; Week 9;n=0,4,2 |  | 1 | 1
  Specific gravity; Week 17;n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  Specific gravity; Week 17;n=0,2,0 |  | 1 |
  Specific gravity; disc/prog;n=0,7,1: number analyzed (Participants) | 0 | 7 | 1
  Specific gravity; disc/prog;n=0,7,1 |  | 2 | 0
  Leukocytes; Week 5;n=1,5,1: number analyzed (Participants) | 1 | 5 | 1
  Leukocytes; Week 5;n=1,5,1 | 0 | 4 | 1
  Leukocytes; Week 9;n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  Leukocytes; Week 9;n=0,1,1 |  | 0 | 1
  Leukocytes; Week 17;n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Leukocytes; Week 17;n=0,1,0 |  | 1 |

22. Primary Outcome: Number of Participants With Maximum Urinalysis Change From Baseline-Part 2
Description: Urine samples were collected for the analysis of following urine parameters: pH, glucose, protein, blood, ketones, specific gravity, erythrocytes and leukocytes. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Only parameters and time points with non-zero values for any increase have been presented.
Time Frame: Baseline (pre-dose Week1 Day1), Weeks 5,9,13,25,37, 49, 73, 85 and discharge/progression
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Participants
  Granular cast;Week5;n=0,2,2,1,3,0: number analyzed (Participants) | 0 | 2 | 2 | 1 | 3 | 0
  Granular cast;Week5;n=0,2,2,1,3,0 |  | 0 | 0 | 0 | 1 |
  Granular cast;disc/prog;n=1,2,6,3,4,0: number analyzed (Participants) | 1 | 2 | 6 | 3 | 4 | 0
  Granular cast;disc/prog;n=1,2,6,3,4,0 | 0 | 0 | 2 | 0 | 0 | 0
  Hyaline cast;Week5;n=1,2,2,2,4,0: number analyzed (Participants) | 1 | 2 | 2 | 2 | 4 | 0
  Hyaline cast;Week5;n=1,2,2,2,4,0 | 1 | 0 | 0 | 1 | 1 |
  Hyaline cast;Week9;n=0,0,1,2,1,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 1
  Hyaline cast;Week9;n=0,0,1,2,1,1 |  |  | 0 | 0 | 0 | 1
  Hyaline cast;Week13;n=1,1,0,0,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  Hyaline cast;Week13;n=1,1,0,0,0,0 | 0 | 1 |  |  |  |
  Hyaline cast;disc/prog;n=1,2,6,3,4,0: number analyzed (Participants) | 1 | 2 | 6 | 3 | 4 | 0
  Hyaline cast;disc/prog;n=1,2,6,3,4,0 | 0 | 0 | 2 | 0 | 0 |
  Glucose;Week 5;n=8,7,18,12,14,8: number analyzed (Participants) | 8 | 7 | 18 | 12 | 14 | 8
  Glucose;Week 5;n=8,7,18,12,14,8 | 1 | 2 | 2 | 0 | 0 | 1
  Glucose;Week9;n=8,3,12,3,6,5: number analyzed (Participants) | 8 | 3 | 12 | 3 | 6 | 5
  Glucose;Week9;n=8,3,12,3,6,5 | 2 | 1 | 0 | 0 | 0 | 0
  Glucose;Week13;n=7,2,6,1,2,2: number analyzed (Participants) | 7 | 2 | 6 | 1 | 2 | 2
  Glucose;Week13;n=7,2,6,1,2,2 | 2 | 1 | 1 | 0 | 0 | 0
  Glucose;Week37;n=3,0,1,0,0,0: number analyzed (Participants) | 3 | 0 | 1 | 0 | 0 | 0
  Glucose;Week37;n=3,0,1,0,0,0 | 1 |  | 0 |  |  |
  Glucose;Week49;n=1,0,1,0,0,0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  Glucose;Week49;n=1,0,1,0,0,0 | 1 |  | 0 |  |  |
  Glucose;Week73;n=1,0,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Glucose;Week73;n=1,0,0,0,0,0 | 1 |  |  |  |  |
  Glucose;Week85;n=1,0,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Glucose;Week85;n=1,0,0,0,0,0 | 1 |  |  |  |  |
  Glucose;disc/prog;n=3,6,16,12,12,5: number analyzed (Participants) | 3 | 6 | 16 | 12 | 12 | 5
  Glucose;disc/prog;n=3,6,16,12,12,5 | 0 | 0 | 0 | 0 | 1 | 0
  Ketones;Week5;n=8,7,18,12,14,8: number analyzed (Participants) | 8 | 7 | 18 | 12 | 14 | 8
  Ketones;Week5;n=8,7,18,12,14,8 | 0 | 1 | 0 | 0 | 1 | 0
  Ketones;Week9;n=8,3,12,3,6,5: number analyzed (Participants) | 8 | 3 | 12 | 3 | 6 | 5
  Ketones;Week9;n=8,3,12,3,6,5 | 0 | 1 | 0 | 0 | 0 | 0
  Ketones;disc/prog;n=3,6,16,12,12,5: number analyzed (Participants) | 3 | 6 | 16 | 12 | 12 | 5
  Ketones;disc/prog;n=3,6,16,12,12,5 | 0 | 1 | 2 | 0 | 1 | 0
  Occult blood;Week5;n=8,7,18,12,14,8: number analyzed (Participants) | 8 | 7 | 18 | 12 | 14 | 8
  Occult blood;Week5;n=8,7,18,12,14,8 | 1 | 0 | 5 | 0 | 0 | 0
  Occult blood;Week9;n=8,3,12,3,6,5: number analyzed (Participants) | 8 | 3 | 12 | 3 | 6 | 5
  Occult blood;Week9;n=8,3,12,3,6,5 | 0 | 1 | 5 | 0 | 0 | 0
  Occult blood;Week13;n=7,2,6,1,2,2: number analyzed (Participants) | 7 | 2 | 6 | 1 | 2 | 2
  Occult blood;Week13;n=7,2,6,1,2,2 | 1 | 0 | 0 | 0 | 0 | 0
  Occult blood;Week25;n=2,0,3,0,0,0: number analyzed (Participants) | 2 | 0 | 3 | 0 | 0 | 0
  Occult blood;Week25;n=2,0,3,0,0,0 | 0 |  | 1 |  |  |
  Occult blood;Week37;n=3,0,1,0,0,0: number analyzed (Participants) | 3 | 0 | 1 | 0 | 0 | 0
  Occult blood;Week37;n=3,0,1,0,0,0 | 1 |  | 0 |  |  |
  Occult blood;disc/prog;n=3,6,16,12,12,5: number analyzed (Participants) | 3 | 6 | 16 | 12 | 12 | 5
  Occult blood;disc/prog;n=3,6,16,12,12,5 | 0 | 0 | 8 | 0 | 0 | 0
  pH;Week5;n=8,7,18,12,14,8: number analyzed (Participants) | 8 | 7 | 18 | 12 | 14 | 8
  pH;Week5;n=8,7,18,12,14,8 | 6 | 3 | 8 | 3 | 6 | 3
  pH;Week9;n=8,3,12,3,6,5: number analyzed (Participants) | 8 | 3 | 12 | 3 | 6 | 5
  pH;Week9;n=8,3,12,3,6,5 | 5 | 1 | 7 | 2 | 4 | 2
  pH;Week13;n=7,2,6,1,2,2: number analyzed (Participants) | 7 | 2 | 6 | 1 | 2 | 2
  pH;Week13;n=7,2,6,1,2,2 | 2 | 1 | 3 | 1 | 0 | 1
  pH;Week25;n=2,0,3,0,0,0: number analyzed (Participants) | 2 | 0 | 3 | 0 | 0 | 0
  pH;Week25;n=2,0,3,0,0,0 | 1 |  | 1 |  |  |
  pH;Week37;n=3,0,1,0,0,0: number analyzed (Participants) | 3 | 0 | 1 | 0 | 0 | 0
  pH;Week37;n=3,0,1,0,0,0 | 3 |  | 0 |  |  |
  pH;Week49;n=1,0,1,0,0,0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  pH;Week49;n=1,0,1,0,0,0 | 1 |  | 0 |  |  |
  pH;Week73;n=1,0,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  pH;Week73;n=1,0,0,0,0,0 | 1 |  |  |  |  |
  pH;Week85;n=1,0,0,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  pH;Week85;n=1,0,0,0,0,0 | 1 |  |  |  |  |
  pH;disc/prog;n=3,6,16,12,12,5: number analyzed (Participants) | 3 | 6 | 16 | 12 | 12 | 5
  pH;disc/prog;n=3,6,16,12,12,5 | 1 | 2 | 6 | 6 | 5 | 2
  Protein;Week5;n=8,7,18,12,14,8: number analyzed (Participants) | 8 | 7 | 18 | 12 | 14 | 8
  Protein;Week5;n=8,7,18,12,14,8 | 1 | 1 | 9 | 3 | 5 | 6
  Protein;Week9;n=8,3,12,3,6,5: number analyzed (Participants) | 8 | 3 | 12 | 3 | 6 | 5
  Protein;Week9;n=8,3,12,3,6,5 | 3 | 2 | 4 | 0 | 0 | 3
  Protein;Week13;n=7,2,6,1,2,2: number analyzed (Participants) | 7 | 2 | 6 | 1 | 2 | 2
  Protein;Week13;n=7,2,6,1,2,2 | 3 | 1 | 2 | 0 | 0 | 0
  Protein;Week37;n=1,0,1,0,0,0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0
  Protein;Week37;n=1,0,1,0,0,0 | 1 |  | 0 |  |  |
  Protein;disc/prog;n=3,6,16,12,12,5: number analyzed (Participants) | 3 | 6 | 16 | 12 | 12 | 5
  Protein;disc/prog;n=3,6,16,12,12,5 | 1 | 1 | 6 | 2 | 3 | 2
  Erythrocytes;Week5;n=3,3,8,4,4,4: number analyzed (Participants) | 3 | 3 | 8 | 4 | 4 | 4
  Erythrocytes;Week5;n=3,3,8,4,4,4 | 2 | 0 | 5 | 2 | 3 | 2
  Erythrocytes;Week9;n=4,0,2,2,1,2: number analyzed (Participants) | 4 | 0 | 2 | 2 | 1 | 2
  Erythrocytes;Week9;n=4,0,2,2,1,2 | 2 |  | 1 | 1 | 1 | 1
  Erythrocytes;Week13;n=3,1,0,0,0,1: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 1
  Erythrocytes;Week13;n=3,1,0,0,0,1 | 3 | 1 |  |  |  | 0
  Erythrocytes;disc/prog;n=1,2,6,3,4,2: number analyzed (Participants) | 1 | 2 | 6 | 3 | 4 | 2
  Erythrocytes;disc/prog;n=1,2,6,3,4,2 | 0 | 0 | 5 | 1 | 2 | 0
  Specific gravity;Week5;n=8,7,18,12,14,8: number analyzed (Participants) | 8 | 7 | 18 | 12 | 14 | 8
  Specific gravity;Week5;n=8,7,18,12,14,8 | 4 | 4 | 2 | 5 | 7 | 2
  Specific gravity;Week9;n=8,3,12,3,6,5: number analyzed (Participants) | 8 | 3 | 12 | 3 | 6 | 5
  Specific gravity;Week9;n=8,3,12,3,6,5 | 2 | 1 | 2 | 2 | 5 | 3
  Specific gravity;Week13;n=7,2,6,1,2,2: number analyzed (Participants) | 7 | 2 | 6 | 1 | 2 | 2
  Specific gravity;Week13;n=7,2,6,1,2,2 | 2 | 1 | 1 | 0 | 0 | 1
  Specific gravity;disc/prog;n=3,6,16,12,12,5: number analyzed (Participants) | 3 | 6 | 16 | 12 | 12 | 5
  Specific gravity;disc/prog;n=3,6,16,12,12,5 | 0 | 2 | 3 | 3 | 5 | 1
  Leukocytes;Week5;n=3,3,8,4,4,4: number analyzed (Participants) | 3 | 3 | 8 | 4 | 4 | 4
  Leukocytes;Week5;n=3,3,8,4,4,4 | 1 | 1 | 5 | 3 | 4 | 4
  Leukocytes;Week9;n=4,0,2,2,1,3: number analyzed (Participants) | 4 | 0 | 2 | 2 | 1 | 3
  Leukocytes;Week9;n=4,0,2,2,1,3 | 0 |  | 2 | 1 | 0 | 3
  Leukocytes;Week13;n=3,1,0,0,0,1: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0 | 1
  Leukocytes;Week13;n=3,1,0,0,0,1 | 1 | 0 |  |  |  | 0
  Leukocytes;Week25;n=2,0,1,0,0,0: number analyzed (Participants) | 2 | 0 | 1 | 0 | 0 | 0
  Leukocytes;Week25;n=2,0,1,0,0,0 | 0 |  | 1 |  |  |
  Leukocytes;disc/prog;n=1,2,7,3,4,1: number analyzed (Participants) | 1 | 2 | 7 | 3 | 4 | 1
  Leukocytes;disc/prog;n=1,2,7,3,4,1 | 0 | 1 | 2 | 3 | 3 | 1

23. Primary Outcome: Number of Participants With Maximum Urinalysis Change From Baseline-Besylate Sub-study
Description: as for outcome 21
Time Frame: Baseline (pre-dose Week1 Day1), Weeks 5,9,17,25 and disc/prog
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  Hyaline casts; Week5;n=1,1: number analyzed (Participants) | 1 | 1
  Hyaline casts; Week5;n=1,1 | 1 | 1
  Hyaline casts; Week9;n=2,1: number analyzed (Participants) | 2 | 1
  Hyaline casts; Week9;n=2,1 | 1 | 0
  Hyaline casts; Week17;n=1,0: number analyzed (Participants) | 1 | 0
  Hyaline casts; Week17;n=1,0 | 1 |
  Hyaline casts; Week25;n=1,0: number analyzed (Participants) | 1 | 0
  Hyaline casts; Week25;n=1,0 | 1 |
  Glucose; Week5;n=3,2: number analyzed (Participants) | 3 | 2
  Glucose; Week5;n=3,2 | 1 | 1
  Glucose; Week9;n=4,1: number analyzed (Participants) | 4 | 1
  Glucose; Week9;n=4,1 | 1 | 0
  Glucose; Week17;n=2,0: number analyzed (Participants) | 2 | 0
  Glucose; Week17;n=2,0 | 1 |
  Ketones; Week9;n=4,1: number analyzed (Participants) | 4 | 1
  Ketones; Week9;n=4,1 | 1 | 0
  pH;Week5;n=3,2: number analyzed (Participants) | 3 | 2
  pH;Week5;n=3,2 | 3 | 1
  pH;Week9;n=4,1: number analyzed (Participants) | 4 | 1
  pH;Week9;n=4,1 | 3 | 0
  pH;Week17;n=2,0: number analyzed (Participants) | 2 | 0
  pH;Week17;n=2,0 | 2 |
  pH;Week25;n=1,0: number analyzed (Participants) | 1 | 0
  pH;Week25;n=1,0 | 1 |
  pH;disc/prog;n=2,2: number analyzed (Participants) | 2 | 2
  pH;disc/prog;n=2,2 | 2 | 1
  Protein; Week5; n=3,2: number analyzed (Participants) | 3 | 2
  Protein; Week5; n=3,2 | 3 | 1
  Protein; Week9; n=4,1: number analyzed (Participants) | 4 | 1
  Protein; Week9; n=4,1 | 3 | 1
  Protein; Week17; n=2,0: number analyzed (Participants) | 2 | 0
  Protein; Week17; n=2,0 | 2 |
  Protein; Week25; n=1,0: number analyzed (Participants) | 1 | 0
  Protein; Week25; n=1,0 | 1 |
  Erythrocytes; Week9; n=4,1: number analyzed (Participants) | 4 | 1
  Erythrocytes; Week9; n=4,1 | 2 | 1
  Erythrocytes; Week17; n=2,0: number analyzed (Participants) | 2 | 0
  Erythrocytes; Week17; n=2,0 | 1 |
  Erythrocytes; Week25; n=1,0: number analyzed (Participants) | 1 | 0
  Erythrocytes; Week25; n=1,0 | 1 |
  Erythrocytes; disc/prog; n=1,0: number analyzed (Participants) | 1 | 0
  Erythrocytes; disc/prog; n=1,0 | 1 |
  Specific gravity; Week5; n=3,2: number analyzed (Participants) | 3 | 2
  Specific gravity; Week5; n=3,2 | 1 | 1
  Specific gravity; Week9; n=4,1: number analyzed (Participants) | 4 | 1
  Specific gravity; Week9; n=4,1 | 2 | 0
  Specific gravity; Week17; n=2,0: number analyzed (Participants) | 2 | 0
  Specific gravity; Week17; n=2,0 | 1 |
  Specific gravity; Week25; n=1,0: number analyzed (Participants) | 1 | 0
  Specific gravity; Week25; n=1,0 | 1 |
  Specific gravity; disc/prog; n=2,2: number analyzed (Participants) | 2 | 2
  Specific gravity; disc/prog; n=2,2 | 0 | 1
  Leukocytes; Week5; n=3,1: number analyzed (Participants) | 3 | 1
  Leukocytes; Week5; n=3,1 | 3 | 1
  Leukocytes; Week9; n=4,1: number analyzed (Participants) | 4 | 1
  Leukocytes; Week9; n=4,1 | 4 | 1
  Leukocytes; Week17; n=2,0: number analyzed (Participants) | 2 | 0
  Leukocytes; Week17; n=2,0 | 1 |
  Leukocytes; Week25; n=1,0: number analyzed (Participants) | 1 | 0
  Leukocytes; Week25; n=1,0 | 1 |
  Leukocytes; disc/prog; n=1,0: number analyzed (Participants) | 1 | 0
  Leukocytes; disc/prog; n=1,0 | 1 |

24. Primary Outcome: Number of Participants With Changes in Pulse Rate From Baseline-Part 1 QD
Description: Pulse rate was measured in a supine or semi-recumbent position after at least 5 minutes rest for the participant. The clinical concern range for pulse rate is <60 beats per minute and >100 beats per minute. Participants were counted twice if the participant "Decreased to <60" and "Increased to >100" post-baseline. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.38 months of drug exposure
Population: All Treated Population. Only those participants with data available at Baseline and the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: GSK525762 2 mg QD: Participants were administered once daily (QD) oral dose of 2 illigrams (mg) GSK525762.
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 8 | 31 | 9
Participants
  Pulse rate; decrease to <60 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
  Pulse rate; Change to normal/no change | 2 | 1 | 0 | 1 | 1 | 5 | 12 | 4
  Pulse rate; increase to >100 | 1 | 2 | 1 | 1 | 3 | 2 | 18 | 5

25. Primary Outcome: Number of Participants With Changes in Pulse Rate From Baseline-Part 1 BID
Description: Pulse rate was measured in a supine or semi-recumbent position after at least 5 minutes rest for the participant. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  Pulse rate; decrease to <60 | 0 | 0 | 0
  Pulse rate; Change to normal/no change | 3 | 4 | 2
  Pulse rate; increase to >100 | 1 | 6 | 3

26. Primary Outcome: Number of Participants With Changes in Pulse Rate From Baseline-Part 2
Description: Pulse rate was measured in a supine or semi-recumbent position after at least 5 minutes rest for the participant. The clinical concern range for pulse rate is <60 beats per minute and >100 beats per minute. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented. Participants were counted twice if the participant "Decreased to <60" and "Increased to >100" post-baseline.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: All Treated Population. Only those participants with data available at Baseline and the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 11 | 14 | 22 | 19 | 20 | 12
Participants
  Pulse rate; decrease to <60 | 0 | 1 | 0 | 0 | 1 | 1
  Pulse rate; Change to normal/no change | 7 | 10 | 13 | 11 | 9 | 8
  Pulse rate; increase to >100 | 5 | 4 | 9 | 9 | 10 | 3

27. Primary Outcome: Number of Participants With Changes in Pulse Rate From Baseline-Besylate Sub-study
Description: Pulse rate was measured in a supine or semi-recumbent position after at least 5 minutes rest for the participant. The clinical concern range for pulse rate is <60 beats per minute and >100 beats per minute. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  Pulse rate; decrease to <60 | 0 | 0
  Pulse rate; Change to normal/no change | 3 | 1
  Pulse rate; increase to >100 | 2 | 4

28. Primary Outcome: Number of Participants With Increase in Blood Pressure From Baseline-Part 1 QD
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) was measured in a supine or semi-recumbent position after at least 5 minutes rest for the participant. Grading of SBP and DBP were done using NCI-CTCAE version 4.0 where, SBP (millimeters of mercury): Grade 0 (<120), Grade 1 (120-139), Grade 2 (140-159), Grade 3/4 (>=160) and DBP: Grade 0 (<80), Grade 1 (80-89), Grade 2 (90-99), Grade 3/4 (>=100). An increase is defined as an increase in CTCAE grade relative to baseline grade. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants
  DBP; Increase to Grade 1 | 2 | 1 | 0 | 0 | 0 | 3 | 9 | 0
  DBP; Increase to Grade 2 | 0 | 0 | 1 | 1 | 1 | 0 | 10 | 1
  DBP; Increase to Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  SBP; Increase to Grade 1 | 1 | 1 | 1 | 1 | 1 | 2 | 11 | 1
  SBP; Increase to Grade 2 | 1 | 0 | 0 | 1 | 3 | 1 | 9 | 3
  SBP; Increase to Grade 3/4 | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 2

29. Primary Outcome: Number of Participants With Increase in Blood Pressure From Baseline-Part 1 BID
Description: SBP and DBP were measured in a supine or semi-recumbent position after at least 5 minutes rest for the participant. Grading of SBP and DBP were done using NCI-CTCAE version 4.0 where, SBP (millimeters of mercury): Grade 0 (<120), Grade 1 (120-139), Grade 2 (140-159), Grade 3/4 (>=160) and DBP: Grade 0 (<80), Grade 1 (80-89), Grade 2 (90-99), Grade 3/4 (>=100). An increase is defined as an increase in CTCAE grade relative to baseline grade. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: All Treated Population. Only those participants with data available at Baseline and the specified time point were analyzed (indicated by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  DBP; Increase to Grade 1;n=4,10,4: number analyzed (Participants) | 4 | 10 | 4
  DBP; Increase to Grade 1;n=4,10,4 | 2 | 4 | 1
  DBP; Increase to Grade 2;n=4,10,4: number analyzed (Participants) | 4 | 10 | 4
  DBP; Increase to Grade 2;n=4,10,4 | 0 | 4 | 1
  DBP; Increase to Grade 3/4;n=4,10,4: number analyzed (Participants) | 4 | 10 | 4
  DBP; Increase to Grade 3/4;n=4,10,4 | 0 | 0 | 1
  SBP; Increase to Grade 1;n=4,9,5: number analyzed (Participants) | 4 | 9 | 5
  SBP; Increase to Grade 1;n=4,9,5 | 1 | 2 | 2
  SBP; Increase to Grade 2;n=4,9,5: number analyzed (Participants) | 4 | 9 | 5
  SBP; Increase to Grade 2;n=4,9,5 | 1 | 6 | 1
  SBP; Increase to Grade 3/4;n=4,9,5: number analyzed (Participants) | 4 | 9 | 5
  SBP; Increase to Grade 3/4;n=4,9,5 | 0 | 0 | 1

30. Primary Outcome: Number of Participants With Changes in Blood Pressure From Baseline-Part 2
Description: as for outcome 29
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: All Treated Population. Only those participants with data available at Baseline and the specified time points were analyzed (indicated by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 11 | 14 | 22 | 19 | 19 | 12
Participants
  DBP; Increase to Grade 1;n=11,14,22,19,19,12 | 2 | 3 | 8 | 5 | 4 | 3
  DBP; Increase to Grade 2;n=11,14,22,19,19,12 | 4 | 1 | 4 | 3 | 6 | 1
  DBP; Increase to Grade 3/4;n=11,14,22,19,19,12 | 0 | 0 | 1 | 2 | 1 | 2
  SBP; Increase to Grade 1;n=11,14,21,19,19,12: number analyzed (Participants) | 11 | 14 | 21 | 19 | 19 | 12
  SBP; Increase to Grade 1;n=11,14,21,19,19,12 | 4 | 4 | 2 | 9 | 7 | 1
  SBP; Increase to Grade 2;n=11,14,21,19,19,12: number analyzed (Participants) | 11 | 14 | 21 | 19 | 19 | 12
  SBP; Increase to Grade 2;n=11,14,21,19,19,12 | 2 | 4 | 11 | 3 | 4 | 7
  SBP; Increase to Grade 3/4;n=11,14,21,19,19,12: number analyzed (Participants) | 11 | 14 | 21 | 19 | 19 | 12
  SBP; Increase to Grade 3/4;n=11,14,21,19,19,12 | 0 | 1 | 3 | 1 | 1 | 0

31. Primary Outcome: Number of Participants With Increase in Blood Pressure From Baseline-Besylate Sub-study
Description: as for outcome 29
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  DBP; Increase to Grade 1 | 1 | 1
  DBP; Increase to Grade 2 | 2 | 1
  DBP; Increase to Grade 3/4 | 0 | 0
  SBP; Increase to Grade 1 | 1 | 1
  SBP; Increase to Grade 2 | 0 | 1
  SBP; Increase to Grade 3/4 | 0 | 0

32. Primary Outcome: Number of Participants With Changes in Temperature From Baseline-Part 1 QD
Description: Temperature was measured in a supine or semi-recumbent position after at least 5 minutes rest for the participant. The clinical concern range for temperature is <=35 degree Celsius and >=38 degree Celsius. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Data for worst case post-Baseline is presented.
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants
  Decrease to <=35 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Change to normal/No change | 3 | 3 | 1 | 3 | 3 | 9 | 27 | 8
  Increase to >=38 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0

33. Primary Outcome: Number of Participants With Changes in Temperature From Baseline-Part 1 BID
Description: as for outcome 32
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  Decrease to <=35 | 0 | 0 | 0
  Change to normal/No change | 4 | 9 | 5
  Increase to >=38 | 0 | 1 | 0

34. Primary Outcome: Number of Participants With Changes in Temperature From Baseline-Part 2
Description: as for outcome 32
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.41 months of drug exposure
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 11 | 14 | 22 | 19 | 20 | 12
Participants
  Decrease to <=35 | 1 | 0 | 0 | 0 | 1 | 0
  Change to normal/No change | 10 | 11 | 20 | 18 | 18 | 12
  Increase to >=38 | 0 | 3 | 2 | 1 | 1 | 0

35. Primary Outcome: Number of Participants With Changes in Temperature From Baseline-Besylate Sub-study
Description: as for outcome 32
Time Frame: Baseline (pre-dose Week1 Day1) and median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  Decrease to <=35 | 0 | 0
  Change to normal/No change | 4 | 5
  Increase to >=38 | 1 | 0

36. Primary Outcome: Overall Response Rate-Part 1 QD
Description: Overall response rate is defined as the percentage of participants who achieved a confirmed complete response (CR) or partial response (PR) from the start of treatment until disease progression or the start of new anticancer therapy, among participants who received at least 1 dose of treatment. Overall response rate was determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST version (v) 1.1). CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeters (mm) in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Percentage of participants | 0 [0.0 to 70.8] | 25 [0.6 to 80.6] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 33.6] | 3 [0.1 to 16.2] | 11 [0.3 to 48.2]

37. Primary Outcome: Overall Response Rate-Part 1 BID
Description: Overall response rate is defined as the percentage of participants who achieved a confirmed CR or PR from the start of treatment until disease progression or the start of new anticancer therapy, among participants who received at least 1 dose of treatment. Overall response rate was determined by the investigator according to RECIST v 1.1. CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Percentage of participants | 0 [0.0 to 60.2] | 0 [0.0 to 30.8] | 0 [0.0 to 52.2]

38. Primary Outcome: Overall Response Rate-Part 2
Description: as for outcome 37
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Percentage of participants | 8 [0.2 to 38.5] | 0 [0.0 to 23.2] | 4 [0.1 to 21.9] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 24.7]

39. Primary Outcome: Overall Response Rate-Besylate Sub-study
Description: as for outcome 37
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population. Data for Besylate sub-study participants were combined for analysis to provide useful interpretation of study data as pre-specified in RAP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants in Besylate Substudy
Number analyzed (Participants) | 10
Percentage of participants | 0 [0.0 to 30.8]

40. Primary Outcome: Number of Participants With Prostate Specific Antigen (PSA)50 Response-Part 1 QD
Description: PSA 50 response rate is defined as the response rate that a PSA reduction from Baseline >=50% is observed at 12 weeks and beyond (must be confirmed by a second value). The number of participants with PSA >=50% reduction is presented along with 95% confidence intervals.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 2 [NA to NA] — Confidence interval could not be calculated as there were no responders | 1 [NA to NA] — Confidence interval could not be calculated as there were no responders

41. Primary Outcome: Number of Participants With PSA50 Response Rate-Part 1 BID
Description: as for outcome 40
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders

42. Primary Outcome: Number of Participants With PSA50 Response-Part 2
Description: as for outcome 40
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Participants | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders

43. Primary Outcome: Number of Participants With PSA50 Response-Besylate Sub-study
Description: as for outcome 40
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders | 0 [NA to NA] — Confidence interval could not be calculated as there were no responders

44. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to 24 Hours(AUC[0 to 24]); AUC From Time 0 to Last Quantifiable Concentration (AUC [0 to t]) and AUC Extrapolated to Infinity (AUC[0 to Inf]) of GSK525762-Besylate Sub-study
Description: Blood samples for pharmacokinetic analysis of GSK525762 were collected at the indicated time points. Besylate sub-study pharmacokinetic (PK) Parameter Population consisted of all participants in the PK Parameter Population who participated in the besylate substudy.
Time Frame: Week1 Day1, Day3 and Week2 Day1 (pre-dose,0.25,0.5,1,1.5,2,3,4,6,8,24,48 hours post-dose)
Population: Besylate Sub-Study PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Groups:
- GSK525762 80 mg Amorphous+6 mg Stable Isotope: Participants were administered GSK525762 80 mg amorphous free-base tablet along with 6 mg stable isotope in the fasted state.
- GSK525762 80 mg Besylate+6 mg Stable Isotope: Participants were administered GSK525762 80 mg besylate tablet along with 6 mg stable isotope in solution in fasted state.
- GSK525762 30 mg Besylate+6 mg Stable Isotope: Participants were administered GSK525762 30 mg besylate tablet along with 6 mg stable isotope in solution in fasted state.
- GSK525762 80 mg Besylate Fed: Participants were administered GSK525762 80 mg besylate tablet along with Food and Drug Administration (FDA) recommended high fat breakfast.
Arm/Group | GSK525762 80 mg Amorphous+6 mg Stable Isotope | GSK525762 80 mg Besylate+6 mg Stable Isotope | GSK525762 30 mg Besylate+6 mg Stable Isotope | GSK525762 80 mg Besylate Fed
Number analyzed (Participants) | 9 | 10 | 10 | 8
Hours*nanograms per milliliter
  AUC(0 to 24) | 6954.3 (59.1) | 7377.9 (44.7) | 2977.3 (42.8) | 9123.8 (45.2)
  AUC(0 to inf) | 7292.0 (62.1) | 7703.4 (49.9) | 3096.9 (45.0) | 9727.7 (48.5)
  AUC(0 to t) | 7227.1 (61.6) | 7657.6 (49.9) | 3053.9 (44.4) | 9597.1 (48.9)

45. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK525762-Besylate Sub-study
Description: Blood samples for pharmacokinetic analysis of GSK525762 were collected at the indicated time points.
Time Frame: Week1 Day1, Day3 and Week2 Day1 (pre-dose,0.25,0.5,1,1.5,2,3,4,6,8,24,48 hours post-dose)
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK525762 80 mg Amorphous+6 mg Stable Isotope | GSK525762 80 mg Besylate+6 mg Stable Isotope | GSK525762 30 mg Besylate+6 mg Stable Isotope | GSK525762 80 mg Besylate Fed
Number analyzed (Participants) | 9 | 10 | 10 | 8
Nanograms per milliliter | 1431.41 (51.3) | 1483.21 (49.8) | 655.33 (21.1) | 1305.59 (46.6)

46. Primary Outcome: Apparent Terminal Phase Elimination Rate Constant (Lambda z) for GSK525762-Besylate Sub-study
Description: Blood samples for pharmacokinetic analysis of GSK525762 were collected at the indicated time points.
Time Frame: Week1 Day1, Day3 and Week2 Day1 (pre-dose,0.25,0.5,1,1.5,2,3,4,6,8,24,48 hours post-dose)
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | GSK525762 80 mg Amorphous+6 mg Stable Isotope | GSK525762 80 mg Besylate+6 mg Stable Isotope | GSK525762 30 mg Besylate+6 mg Stable Isotope | GSK525762 80 mg Besylate Fed
Number analyzed (Participants) | 9 | 10 | 10 | 8
Per hour | 5.628 (25.9) | 5.176 (20.6) | 5.088 (23.8) | 5.954 (20.2)

47. Primary Outcome: Time to Reach Cmax (Tmax) for GSK525762-Besylate Sub-study
Description: Blood samples for pharmacokinetic analysis of GSK525762 were collected at the indicated time points.
Time Frame: Week1 Day1, Day3 and Week2 Day1 (pre-dose,0.25,0.5,1,1.5,2,3,4,6,8,24,48 hours post-dose)
Population: as for outcome 44
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK525762 80 mg Amorphous+6 mg Stable Isotope | GSK525762 80 mg Besylate+6 mg Stable Isotope | GSK525762 30 mg Besylate+6 mg Stable Isotope | GSK525762 80 mg Besylate Fed
Number analyzed (Participants) | 9 | 10 | 10 | 8
Hours | 0.5833 [0.250 to 3.250] | 0.8083 [0.500 to 3.000] | 0.8333 [0.300 to 1.017] | 2.0000 [0.500 to 6.050]

48. Secondary Outcome: Number of Participants With Increase in QT Interval Corrected for Heart Rate According to Fridericia's Formula (QTcF)-Part 1 QD
Description: Electrocardiogram (ECG) measurements were done using an automated 12-lead ECG machine. QTc parameters were graded according to NCI-CTCAE version 4.0. Grade 0 (<450 milliseconds [msec]), Grade 1 (450-480 msec), Grade 2 (481-500 msec), Grade 3 (>=501 msec). An increase is defined as an increase in CTCAE grade relative to Baseline grade. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Number of participants with increase in QTcF at worst-case post Baseline is reported.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Participants
  Any Grade increase | 1 | 0 | 0 | 1 | 4 | 4 | 13 | 4
  Increase to Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Increase to Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Number of Participants With Increase in QTcF-Part 1 BID
Description: ECG measurements were done using an automated 12-lead ECG machine. QTc parameters were graded according to NCI-CTCAE version 4.0. Grade 0 (<450 milliseconds [msec]), Grade 1 (450-480 msec), Grade 2 (481-500 msec), Grade 3 (>=501 msec). An increase is defined as an increase in CTCAE grade relative to Baseline grade. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Number of participants with increase in QTcF at worst-case post Baseline is reported.
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Participants
  Any Grade increase | 3 | 4 | 2
  Increase to Grade 2 | 3 | 0 | 0
  Increase to Grade 3 | 0 | 0 | 0

50. Secondary Outcome: Number of Participants With Increase in QTcF-Part 2
Description: as for outcome 49
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 11 | 14 | 22 | 19 | 20 | 12
Participants
  Any Grade increase | 1 | 2 | 6 | 1 | 2 | 0
  Increase to Grade 2 | 0 | 0 | 0 | 0 | 2 | 0
  Increase to Grade 3 | 1 | 0 | 0 | 0 | 0 | 0

51. Secondary Outcome: Number of Participants With Increase in QTcF-Besylate Sub-study
Description: ECG measurements were done using 12-lead ECG machine that automatically calculated the heart rate and measured PR, QRS, QT and QTcF intervals. QTc parameters were graded according to NCI-CTCAE version 4.0. Grade 0 (<450 milliseconds [msec]), Grade 1 (450-480 msec), Grade 2 (481-500 msec), Grade 3 (>=501 msec). An increase is defined as an increase in CTCAE grade relative to Baseline grade. Baseline is the most recent, non-missing value prior to or on the first study treatment dose date. Number of participants with increase in QTcF at worst-case post Baseline is reported.
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  Any Grade increase | 2 | 0
  Increase to Grade 2 | 0 | 0
  Increase to Grade 3 | 0 | 0

52. Secondary Outcome: Progression Free Survival-Part 1 QD
Description: Progression free survival is defined as the interval of time (in months) between the date of first dose and the earlier of the date of disease progression and date of death due to any cause. Confidence intervals were estimated using Brookmeyer Crowley method.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Months | 0.3 [0.3 to 0.4] | 4.1 [0.9 to 13.9] | 2.2 [NA to NA] — Confidence interval could not be calculated as only one participant was analyzed | 9.1 [1.4 to 13.9] | 3.8 [0.9 to 5.4] | 3.6 [1.4 to 8.9] | 6.5 [2.6 to 9.1] | 7.5 [6.0 to 18.0]

53. Secondary Outcome: Progression Free Survival-Part 1 BID
Description: as for outcome 52
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Months | 7.7 [0.9 to 14.5] | 5.6 [2.9 to 7.0] | 8.0 [7.9 to 18.7]

54. Secondary Outcome: Progression Free Survival-Part 2
Description: Progression free survival is defined as the interval of time (in months) between the date of first dose and the earlier of the date of disease progression and the date of death due to any cause. Confidence intervals were estimated using Brookmeyer Crowley method.
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Months | 4.8 [2.5 to 5.1] | 2.2 [1.1 to 5.3] | 8.0 [5.5 to 11.7] | 2.4 [1.4 to 6.5] | 4.7 [3.3 to 9.2] | 3.4 [1.9 to 7.3]

55. Secondary Outcome: Progression Free Survival-Besylate Sub-study
Description: as for outcome 54
Time Frame: Median of 1.87 months of drug exposure
Population: as for outcome 39
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants in Besylate Substudy
Number analyzed (Participants) | 10
Months | 3.5 [1.0 to 10.9]

56. Secondary Outcome: Time to Response-Part 1 QD
Description: Time to response is defined, for participants with a confirmed CR or PR, as the time from first dose to the first documented evidence of CR or PR. Time to response is not derived for participants with incomplete response dates. Confidence intervals were estimated using Brookmeyer Crowley method.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Groups:
- Part 1: GSK525762 2 mg QD: Participants were administered once daily (QD) oral dose of 2 milligrams(mg) GSK525762
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Time to Response-Part 1 BID
Description: as for outcome 56
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 0 | 0 | 0

58. Secondary Outcome: Time to Response-Part 2
Description: as for outcome 56
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

59. Secondary Outcome: Time to Response-Besylate Sub-study
Description: as for outcome 56
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 0 | 0

60. Secondary Outcome: Duration of Response-Part 1 QD
Description: Duration of response is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause among participants who achieve a confirmed CR or PR. Duration of response is not derived for participants with incomplete response dates. Confidence intervals were estimated using Brookmeyer Crowley method.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

61. Secondary Outcome: Duration of Response-Part 1 BID
Description: as for outcome 60
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 0 | 0 | 0

62. Secondary Outcome: Duration of Response-Part 2
Description: as for outcome 60
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

63. Secondary Outcome: Duration of Response-Besylate Sub-study
Description: as for outcome 60
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population. Participants with incomplete response dates were excluded from the analysis.
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Overall Survival-Part 1 QD
Description: Overall survival is defined as the interval of time (in months) between the date of first dose and the date of death due to any cause. The median overall survival is presented along with 95% confidence interval. Confidence intervals were estimated using Brookmeyer Crowley method.
Time Frame: Median of 1.38 months of drug exposure
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Months | 0.6 [0.3 to NA] — The upper limit of the 95% CI could not be estimated due to the low number of participants being analyzed. | 4.1 [0.9 to 13.9] | 2.2 [NA to NA] — Confidence interval could not be calculated as only one participant was analyzed | 9.1 [5.6 to 13.9] | 3.8 [2.8 to 5.4] | 8.9 [3.6 to 20.2] | 7.1 [3.9 to 9.5] | 9.8 [6.0 to 18.0]

65. Secondary Outcome: Overall Survival-Part 1 BID
Description: as for outcome 64
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Months | NA [14.5 to NA] — Values could not be estimated due to limited amount of observed follow-up time. | 6.0 [2.9 to 12.2] | 13.3 [7.9 to 18.7]

66. Secondary Outcome: Overall Survival-Part 2
Description: as for outcome 64
Time Frame: Median of 1.41 months of drug exposure
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants With NMC | Participants With SCLC | Participants With CRPC | Participants With TNBC | Participants With ER+BC | Participants With GIST
Number analyzed (Participants) | 12 | 14 | 23 | 19 | 21 | 13
Months | 5.0 [4.3 to NA] — The upper limit of the 95% CI could not be estimated due to the low number of participants being analyzed. | 2.6 [1.1 to 9.4] | 9.1 [6.7 to 11.7] | 5.0 [2.3 to 10.3] | 8.8 [3.6 to 13.1] | 7.3 [3.4 to NA] — The upper limit of the 95% CI could not be estimated due to the low number of participants being analyzed.

67. Secondary Outcome: Overall Survival-Besylate Sub-study
Description: as for outcome 64
Time Frame: Median of 1.87 months of drug exposure
Population: as for outcome 39
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants in Besylate Substudy
Number analyzed (Participants) | 10
Months | 6.3 [3.6 to 10.9]

68. Secondary Outcome: AUC (0 to t), AUC (0 to 24) and AUC (0 to Inf) of GSK525762-Part 1 QD
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK525762. PK parameter population comprised of all participants in the PK Concentration Population (all participants in the All Treated Population for whom a blood sample for pharmacokinetics is obtained and analyzed) for whom a PK parameter has been obtained.
Time Frame: pre-dose,0.25,0.5,1,2,4,8,12,24 and 48 hours post-dose at Week1 Day1 and Week 3 Day 4
Population: PK Parameter Population. Only those participants with data available at the specified time points were available (indicated by n=X in category titles)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Part 1: GSK525762 2 mg QD: Participants were administered once daily oral dose of 2 mg GSK525762.
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Hours*nanogram per milliliter
  AUC (0 to 24); Week1;n=3,4,1,3,4,9,32,9 | 169.2 (39.4) | 354.3 (33.8) | 431.5 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 867.9 (39.5) | 3943.2 (49.5) | 4225.0 (39.2) | 5692.4 (61.4) | 6958.3 (43.5)
  AUC (0 to 24); Week3;n=1,2,1,3,4,6,16,6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 4 | 6 | 16 | 6
  AUC (0 to 24); Week3;n=1,2,1,3,4,6,16,6 | 152.9 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 334.6 (60.5) | 329.5 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 671.6 (21.4) | 3146.2 (54.5) | 2575.6 (47.3) | 2959.8 (48.4) | 3818.5 (35.8)
  AUC (0 to inf); Week1;n=3,4,1,3,4,9,32,9 | 174.4 (44.3) | 360.8 (35.1) | 433.1 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 887.1 (39.1) | 4464.5 (62.9) | 4357.5 (42.1) | 5887.2 (62.8) | 7295.6 (45.2)
  AUC (0 to t); Week1;n=3,4,1,3,4,9,32,9 | 168.6 (44.5) | 357.5 (34.8) | 431.1 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 877.7 (39.4) | 4147.8 (54.3) | 4304.1 (40.7) | 5667.3 (61.5) | 7218.4 (45.1)
  AUC (0 to t); Week3;n=1,2,1,3,4,6,16,6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 4 | 6 | 16 | 6
  AUC (0 to t); Week3;n=1,2,1,3,4,6,16,6 | 152.8 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 334.3 (60.3) | 330.6 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 672.3 (21.5) | 3164.3 (54.7) | 2576.9 (47.3) | 2953.8 (49.0) | 3819.9 (35.9)

69. Secondary Outcome: Maximum Observed Concentration for GSK525762-Part 1 QD
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK525762.
Time Frame: pre-dose,0.25,0.5,1,2,4,8,12,24 and 48 hours post-dose at Week1 Day1 and Week 3 Day 4
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Nanogram per milliliter
  Week1;n=3,4,1,3,4,9,32,9 | 50.95 (41.5) | 70.46 (29.2) | 120.35 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 179.45 (39.9) | 603.92 (30.3) | 889.52 (24.5) | 1099.81 (62.7) | 1080.49 (38.8)
  Week3;n=1,2,1,3,4,6,16,6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 4 | 6 | 16 | 6
  Week3;n=1,2,1,3,4,6,16,6 | 52.04 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 53.37 (16.3) | 103.18 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 137.57 (25.1) | 602.70 (17.2) | 633.71 (52.6) | 815.40 (41.1) | 918.56 (41.4)

70. Secondary Outcome: Lambda z for GSK525762-Part 1 QD
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK525762.
Time Frame: pre-dose,0.25,0.5,1,2,4,8,12,24 and 48 hours post-dose at Week1 Day1 and Week 3 Day 4
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Per hour
  Week1;n=3,4,1,3,4,9,32,9 | 0.21411 (98.4) | 0.13554 (37.4) | 0.23126 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 0.09903 (43.5) | 0.07863 (53.1) | 0.12468 (28.2) | 0.15613 (34.1) | 0.10992 (16.0)
  Week3;n=1,2,1,3,4,6,16,6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 4 | 6 | 16 | 6
  Week3;n=1,2,1,3,4,6,16,6 | 0.15579 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 0.15472 (11.2) | 0.14087 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 0.15599 (21.7) | 0.12513 (12.7) | 0.17629 (26.3) | 0.16667 (30.6) | 0.17560 (21.1)

71. Secondary Outcome: Tmax for GSK525762-Part 1 QD
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK525762.
Time Frame: pre-dose,0.25,0.5,1,2,4,8,12,24 and 48 hours post-dose at Week1 Day1 and Week 3 Day 4
Population: as for outcome 69
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Hours
  Week1;n=3,4,1,3,4,9,32,9 | 0.5833 [0.500 to 0.633] | 1.2250 [0.500 to 2.000] | 1.1000 [1.100 to 1.100] | 2.0167 [0.333 to 3.967] | 2.0083 [0.967 to 2.233] | 1.0000 [0.517 to 4.000] | 1.0000 [0.250 to 4.000] | 1.0000 [0.667 to 3.950]
  Week3;n=1,2,1,3,4,6,16,6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 4 | 6 | 16 | 6
  Week3;n=1,2,1,3,4,6,16,6 | 1.0000 [1.000 to 1.000] | 2.5083 [1.017 to 4.000] | 0.5000 [0.500 to 0.500] | 1.0500 [0.767 to 4.000] | 0.9000 [0.317 to 4.000] | 1.0583 [0.500 to 2.033] | 0.5667 [0.300 to 4.017] | 1.5000 [0.500 to 2.000]

72. Secondary Outcome: Apparent Clearance of GSK525762-Part 1 QD
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK525762.
Time Frame: pre-dose,0.25,0.5,1,2,4,8,12,24 and 48 hours post-dose at Week1 Day1 and Week 3 Day 4
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Liter per hour
  Week1;n=3,4,1,3,4,9,32,9 | 11.467 (44.3) | 11.085 (35.1) | 18.470 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 18.036 (39.1) | 6.720 (62.9) | 13.769 (42.1) | 13.589 (62.8) | 13.707 (45.2)
  Week3;n=1,2,1,3,4,6,16,6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 4 | 6 | 16 | 6
  Week3;n=1,2,1,3,4,6,16,6 | 13.082 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 11.955 (60.5) | 24.277 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 23.823 (21.4) | 9.535 (54.5) | 23.296 (47.3) | 27.029 (48.4) | 26.188 (35.8)

73. Secondary Outcome: Volume of Distribution of GSK525762-Part 1 QD
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK525762.
Time Frame: pre-dose,0.25,0.5,1,2,4,8,12,24 and 48 hours post-dose at Week1 Day1 and Week 3 Day 4
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: GSK525762 2 mg QD | Part 1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 9 | 32 | 9
Liters
  Week1;n=3,4,1,3,4,9,32,9 | 53.56 (65.9) | 81.79 (34.7) | 79.87 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 182.13 (92.7) | 85.46 (30.3) | 110.44 (23.5) | 87.03 (56.4) | 124.70 (42.6)
  Week3;n=1,2,1,3,4,6,16,6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 4 | 6 | 16 | 6
  Week3;n=1,2,1,3,4,6,16,6 | 83.97 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 77.27 (47.0) | 172.33 (NA) — Geometric coefficient of variation could not be calculated as only one participant was analyzed at the specified time point. | 152.72 (44.5) | 76.20 (44.0) | 132.14 (34.7) | 162.17 (40.6) | 149.14 (26.9)

74. Secondary Outcome: AUC (0 to Inf), AUC (0 to 24) and AUC (0 to t) of GSK525762-Part 1 BID
Description: Blood samples were collected at indicated time points post ante-meridiem (AM) and post-meridiem (PM) dose for pharmacokinetic analysis of GSK525762.
Time Frame: pre-dose,0.25,0.5,1,2,4,8,12 hours post-AM dose at Week1Day1 and Week3 Day 4; Week1 Day5(0.5, 3 hours post-AM dose); pre-dose, 0.25,0.5,1,2,4,8,12, 36 hours post-PM dose at Week1Day1 and Week3 Day4
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliter
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Hours*nanogram per milliter
  AUC (0 to 24); Week1 AM dose;n=3,10,5: number analyzed (Participants) | 3 | 10 | 5
  AUC (0 to 24); Week1 AM dose;n=3,10,5 | 856.1 (123.7) | 3067.0 (43.9) | 2794.4 (31.8)
  AUC (0 to 24); Week1 PM dose;n=4,7,5: number analyzed (Participants) | 4 | 7 | 5
  AUC (0 to 24); Week1 PM dose;n=4,7,5 | 981.4 (84.8) | 3261.1 (59.9) | 2607.6 (36.2)
  AUC (0 to 24); Week3 AM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  AUC (0 to 24); Week3 AM dose;n=3,7,3 | 1279.0 (116.2) | 2725.3 (92.4) | 1184.6 (17.8)
  AUC (0 to 24); Week3 PM dose;n=3,5,3: number analyzed (Participants) | 3 | 5 | 3
  AUC (0 to 24); Week3 PM dose;n=3,5,3 | 1155.8 (102.4) | 1662.1 (29.2) | 1131.6 (28.5)
  AUC (0 to inf); Week1 AM dose;n=3,10,5: number analyzed (Participants) | 3 | 10 | 5
  AUC (0 to inf); Week1 AM dose;n=3,10,5 | 860.4 (124.4) | 3118.3 (45.3) | 2825.8 (32.8)
  AUC (0 to t); Week1 AM dose;n=4,10,5 | 932.2 (97.6) | 2727.2 (40.8) | 2579.0 (28.0)
  AUC (0 to t); Week1 PM dose;n=4,9,5: number analyzed (Participants) | 4 | 9 | 5
  AUC (0 to t); Week1 PM dose;n=4,9,5 | 927.5 (82.5) | 2840.4 (43.4) | 2446.7 (34.2)
  AUC (0 to t); Week3 AM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  AUC (0 to t); Week3 AM dose;n=3,7,3 | 1194.6 (110.1) | 2472.4 (89.8) | 1140.9 (16.9)
  AUC (0 to t); Week3 PM dose;n=3,6,3: number analyzed (Participants) | 3 | 6 | 3
  AUC (0 to t); Week3 PM dose;n=3,6,3 | 1053.6 (96.6) | 1490.8 (23.3) | 1073.6 (29.2)

75. Secondary Outcome: Maximum Observed Concentration of GSK525762-Part 1 BID
Description: as for outcome 74
Time Frame: as for outcome 74
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliter
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Nanogram per milliter
  Week1 AM dose;n=4,10,5 | 231.68 (70.6) | 628.01 (40.0) | 703.31 (34.2)
  Week1 PM dose;n=4,9,5: number analyzed (Participants) | 4 | 9 | 5
  Week1 PM dose;n=4,9,5 | 166.62 (62.0) | 445.17 (27.6) | 425.76 (29.3)
  Week3 AM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Week3 AM dose;n=3,7,3 | 284.71 (87.1) | 604.38 (66.4) | 419.15 (18.1)
  Week3 PM dose;n=3,6,3: number analyzed (Participants) | 3 | 6 | 3
  Week3 PM dose;n=3,6,3 | 256.08 (94.0) | 263.72 (41.3) | 229.91 (34.8)

76. Secondary Outcome: Lambda z for GSK525762-Part 1 BID
Description: as for outcome 74
Time Frame: as for outcome 74
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Per hour
  Week1 AM dose;n=3,10,5: number analyzed (Participants) | 3 | 10 | 5
  Week1 AM dose;n=3,10,5 | 0.23463 (19.4) | 0.19989 (29.6) | 0.23721 (39.4)
  Week1 PM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Week1 PM dose;n=3,7,3 | 0.21171 (23.1) | 0.14307 (36.6) | 0.18789 (25.2)
  Week3 AM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Week3 AM dose;n=3,7,3 | 0.23565 (27.2) | 0.21751 (27.7) | 0.30868 (19.6)
  Week3 PM dose;n=3,5,3: number analyzed (Participants) | 3 | 5 | 3
  Week3 PM dose;n=3,5,3 | 0.20507 (21.5) | 0.19263 (27.7) | 0.29133 (15.8)

77. Secondary Outcome: Tmax for GSK525762-Part 1 BID
Description: as for outcome 74
Time Frame: as for outcome 74
Population: as for outcome 69
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Hour
  Week1 AM dose;n=4,10,5 | 1.5500 [0.583 to 4.283] | 0.9667 [0.550 to 2.100] | 0.5500 [0.517 to 1.033]
  Week1 PM dose;n=4,9,5: number analyzed (Participants) | 4 | 9 | 5
  Week1 PM dose;n=4,9,5 | 1.9583 [1.917 to 4.000] | 1.9667 [0.967 to 4.167] | 1.9833 [1.017 to 7.733]
  Week3 AM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Week3 AM dose;n=3,7,3 | 1.1833 [1.167 to 2.067] | 1.0667 [0.250 to 2.017] | 0.5833 [0.183 to 1.000]
  Week3 PM dose;n=3,6,3: number analyzed (Participants) | 3 | 6 | 3
  Week3 PM dose;n=3,6,3 | 1.0000 [0.500 to 2.083] | 1.4500 [0.000 to 2.083] | 2.0667 [1.900 to 2.067]

78. Secondary Outcome: Apparent Clearance of GSK525762-Part 1 BID
Description: as for outcome 74
Time Frame: as for outcome 74
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Liter per hour
  Week1 AM dose;n=3,10,5: number analyzed (Participants) | 3 | 10 | 5
  Week1 AM dose;n=3,10,5 | 23.246 (124.4) | 9.621 (45.3) | 14.155 (32.8)
  Week1 PM dose;n=4,7,5: number analyzed (Participants) | 4 | 7 | 5
  Week1 PM dose;n=4,7,5 | 21.745 (82.7) | 11.057 (48.1) | 16.382 (34.6)
  Week3 AM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Week3 AM dose;n=3,7,3 | 16.731 (110.1) | 11.949 (86.1) | 34.623 (18.7)
  Week3 PM dose;n=3,5,3: number analyzed (Participants) | 3 | 5 | 3
  Week3 PM dose;n=3,5,3 | 18.867 (96.0) | 20.133 (26.2) | 37.097 (29.4)

79. Secondary Outcome: Volume of Distribution of GSK525762-Part 1 BID
Description: as for outcome 74
Time Frame: as for outcome 74
Population: as for outcome 69
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID
Number analyzed (Participants) | 4 | 10 | 5
Liters
  Week1 AM dose;n=3,10,5: number analyzed (Participants) | 3 | 10 | 5
  Week1 AM dose;n=3,10,5 | 99.07 (91.0) | 48.13 (40.8) | 59.67 (35.0)
  Week1 PM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Week1 PM dose;n=3,7,3 | 116.52 (66.0) | 77.28 (16.6) | 81.11 (52.6)
  Week3 AM dose;n=3,7,3: number analyzed (Participants) | 3 | 7 | 3
  Week3 AM dose;n=3,7,3 | 71.00 (72.8) | 54.94 (61.4) | 112.17 (37.6)
  Week3 PM dose;n=3,5,3: number analyzed (Participants) | 3 | 5 | 3
  Week3 PM dose;n=3,5,3 | 92.00 (65.3) | 104.52 (29.5) | 127.34 (41.7)

80. Primary Outcome: Number of Participants With Non-serious AEs and SAEs-Besylate Sub-study
Description: as for outcome 2
Time Frame: Median of 1.87 months of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | 80mg Amor+6mg Iso/80mg Bes+6mg Iso/30mg Bes+6mg Iso/80mg Bes | 80mg Bes+6mg Iso/80mg Amor+6mg Iso/30mg Bes+6mg Iso/80mg Bes
Number analyzed (Participants) | 5 | 5
Participants
  Any non-serious AE | 5 | 5
  Any SAE | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from the start of study treatment until 28 days following discontinuation of study treatment (Median of 1.38 months of drug exposure-Part 1 QD, Median of 1.41 months of drug exposure-Part 1 BID and Part 2 and Median of 1.87 months of drug exposure-Besylate sub-study).
Description: Adverse events were collected in the All Treated Population.
Groups:
- Part1: GSK525762 4 mg QD: Participants were administered once daily oral dose of 4 mg GSK525762.
- Part1: GSK525762 2 mg QD: Participants were administered once daily (QD) oral dose of 2 milligrams (mg) GSK525762.
- 80mg Amor+6mg Iso/80mg Bes+6mg: Participants received GSK525762 80 mg amorphous (amor) free-base tablet along with 6 mg stable isotope (iso) in solution in the fasted state in Period 1 followed by administration of GSK525762 80 mg besylate (bes) tablet along with 6 mg stable iso in solution in the fasted state in Period 2. Participants were then administered GSK525762 30 mg bes tablet along with 6 mg stable iso in solution in the fasted state in Period 3 and GSK525762 80 mg bes tablet was administered with Food and Drug Administration (FDA) recommended high fat breakfast in Period 4.
- 80mg Bes+6mg Iso/80mg Amor+6mg: Participants received GSK525762 80 mg bes tablet along with 6 mg stable iso in solution in the fasted state in Period 1 followed by administration GSK525762 80 mg amor free-base tablet along with 6 mg stable iso in solution in the fasted state in Period 2. Participants were then administered GSK525762 30 mg bes tablet along with 6 mg stable iso in solution in the fasted state in Period 3 and GSK525762 80 mg bes tablet was administered with FDA recommended high fat breakfast in Period 4.
Arm/Group | Part1: GSK525762 4 mg QD | Part 1: GSK525762 8 mg QD | Part 1: GSK525762 16 mg QD | Part 1: GSK525762 30 mg QD | Part 1: GSK525762 60 mg QD | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 100 mg QD | Part 1: GSK525762 20 mg BID | Part 1: GSK525762 30 mg BID | Part 1: GSK525762 40 mg BID | Part 2: Participants With NMC | Part 2: Participants With SCLC | Part 2: Participants With CRPC | Part1: GSK525762 2 mg QD | Part 2: Participants With TNBC | Part 2: Participants With ER+BC | Part 2: Participants With GIST | 80mg Amor+6mg Iso/80mg Bes+6mg | 80mg Bes+6mg Iso/80mg Amor+6mg
All-Cause Mortality (participants affected / at risk) | 4/4 | 1/1 | 3/3 | 4/4 | 7/9 | 30/32 | 7/9 | 1/4 | 9/10 | 3/5 | 8/12 | 12/14 | 21/23 | 2/3 | 16/19 | 17/21 | 5/13 | 1/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/1 | 0/3 | 1/4 | 2/9 | 21/32 | 3/9 | 0/4 | 4/10 | 2/5 | 6/12 | 9/14 | 16/23 | 0/3 | 11/19 | 15/21 | 8/13 | 3/5 | 3/5
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1 | 3/3 | 3/4 | 9/9 | 31/32 | 9/9 | 4/4 | 10/10 | 5/5 | 11/12 | 14/14 | 23/23 | 3/3 | 19/19 | 21/21 | 12/13 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1: GSK525762 4 mg QD (N=4) | Part 1: GSK525762 8 mg QD (N=1) | Part 1: GSK525762 16 mg QD (N=3) | Part 1: GSK525762 30 mg QD (N=4) | Part 1: GSK525762 60 mg QD (N=9) | Part 1: GSK525762 80 mg QD (N=32) | Part 1: GSK525762 100 mg QD (N=9) | Part 1: GSK525762 20 mg BID (N=4) | Part 1: GSK525762 30 mg BID (N=10) | Part 1: GSK525762 40 mg BID (N=5) | Part 2: Participants With NMC (N=12) | Part 2: Participants With SCLC (N=14) | Part 2: Participants With CRPC (N=23) | Part1: GSK525762 2 mg QD (N=3) | Part 2: Participants With TNBC (N=19) | Part 2: Participants With ER+BC (N=21) | Part 2: Participants With GIST (N=13) | 80mg Amor+6mg Iso/80mg Bes+6mg (N=5) | 80mg Bes+6mg Iso/80mg Amor+6mg (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiotoxicity (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulation factor VII level decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (10) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 4 (5) | 9 (10) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyrotoxic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1: GSK525762 4 mg QD (N=4) | Part 1: GSK525762 8 mg QD (N=1) | Part 1: GSK525762 16 mg QD (N=3) | Part 1: GSK525762 30 mg QD (N=4) | Part 1: GSK525762 60 mg QD (N=9) | Part 1: GSK525762 80 mg QD (N=32) | Part 1: GSK525762 100 mg QD (N=9) | Part 1: GSK525762 20 mg BID (N=4) | Part 1: GSK525762 30 mg BID (N=10) | Part 1: GSK525762 40 mg BID (N=5) | Part 2: Participants With NMC (N=12) | Part 2: Participants With SCLC (N=14) | Part 2: Participants With CRPC (N=23) | Part1: GSK525762 2 mg QD (N=3) | Part 2: Participants With TNBC (N=19) | Part 2: Participants With ER+BC (N=21) | Part 2: Participants With GIST (N=13) | 80mg Amor+6mg Iso/80mg Bes+6mg (N=5) | 80mg Bes+6mg Iso/80mg Amor+6mg (N=5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 2 (2) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 4 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 11 (14) | 5 (5) | 2 (2) | 4 (4) | 1 (2) | 3 (3) | 6 (6) | 13 (14) | 0 (0) | 7 (7) | 9 (11) | 2 (2) | 4 (4) | 3 (3)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anhedonia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 6 (8) | 0 (0) | 4 (4) | 6 (7) | 2 (2) | 2 (6) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 0 (0) | 1 (1) | 7 (8) | 3 (4) | 5 (6) | 4 (5) | 6 (6) | 0 (0) | 7 (9) | 11 (12) | 3 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (6) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood insulin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coagulation factor VII level decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 3 (3) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 5 (6) | 1 (2) | 2 (2) | 4 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 15 (19) | 6 (8) | 1 (1) | 7 (10) | 4 (5) | 4 (4) | 5 (5) | 15 (16) | 0 (0) | 8 (8) | 10 (11) | 6 (6) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 11 (16) | 4 (5) | 0 (0) | 6 (10) | 5 (8) | 6 (8) | 4 (6) | 12 (24) | 1 (1) | 7 (7) | 8 (11) | 4 (5) | 3 (5) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 8 (9) | 5 (6) | 1 (1) | 4 (4) | 2 (2) | 4 (4) | 2 (2) | 10 (12) | 0 (0) | 5 (6) | 7 (8) | 5 (5) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 5 (6) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 4 (4) | 5 (5) | 0 (0) | 4 (4) | 8 (8) | 4 (4) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Factor V deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 11 (12) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 5 (5) | 12 (15) | 1 (1) | 7 (7) | 4 (4) | 3 (3) | 3 (3) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (11) | 5 (6) | 1 (1) | 4 (4) | 2 (3) | 6 (8) | 4 (5) | 7 (9) | 0 (0) | 2 (3) | 9 (12) | 2 (2) | 2 (2) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 4 (7) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 6 (7) | 5 (5) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 5 (5) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 4 (4) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 2 (2) | 15 (19) | 7 (10) | 2 (2) | 6 (9) | 1 (2) | 5 (6) | 8 (8) | 11 (16) | 0 (0) | 8 (12) | 9 (12) | 5 (5) | 3 (4) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 2 (3) | 4 (7) | 4 (4) | 1 (1) | 2 (2)
Prothrombin time ratio decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 5 (5) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 18 (39) | 5 (8) | 1 (1) | 7 (8) | 5 (5) | 3 (5) | 7 (12) | 12 (23) | 0 (0) | 13 (15) | 13 (18) | 3 (3) | 4 (4) | 3 (3)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 11 (20) | 4 (5) | 3 (3) | 3 (6) | 1 (1) | 4 (5) | 4 (4) | 9 (18) | 0 (0) | 8 (11) | 6 (8) | 2 (2) | 3 (3) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 0 (0) | 3 (4) | 1 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT01587703/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT01587703/SAP_001.pdf